CLINICAL TRIAL: NCT03329092
Title: A PHASE 3 PROSPECTIVE, RANDOMIZED, MULTICENTER, OPEN-LABEL, CENTRAL ASSESSOR-BLINDED, PARALLEL GROUP, COMPARATIVE STUDY TO DETERMINE THE EFFICACY, SAFETY AND TOLERABILITY OF AZTREONAM-AVIBACTAM (ATM-AVI) ±METRONIDAZOLE (MTZ) VERSUS MEROPENEM±COLISTIN (MER±COL) FOR THE TREATMENT OF SERIOUS INFECTIONS DUE TO GRAM NEGATIVE BACTERIA, INCLUDING METALLO-Β-LACTAMASE (MBL) - PRODUCING MULTIDRUG RESISTANT PATHOGENS, FOR WHICH THERE ARE LIMITED OR NO TREATMENT OPTIONS
Brief Title: A Study to Determine the Efficacy, Safety and Tolerability of Aztreonam-Avibactam (ATM-AVI) ± Metronidazole (MTZ) Versus Meropenem (MER) ± Colistin (COL) for the Treatment of Serious Infections Due to Gram Negative Bacteria.
Acronym: REVISIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Innovative Medicines Initiative (Other); Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C3601002; D4910C00004 (Other: Alias Study Number); 2017-002742-68 (EudraCT Number)
Record Dates: First submitted 2017-10-06; First posted 2017-11-01 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Complicated Intra-abdominal Infection; Hosptial Acquired Pneumonia; Ventilator Associated Pneumonia
Keywords: Complicated intra-abdominal infection; Hosptial acquired pneumonia; Ventilator associated pneumonia; Gram negative infections; Metallo-beta lactamase; Multi drug resistant pathogens
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Multicenter, Open Label, Central Assessor Blinded, Parallel Group, Comparative Study
Who Masked: Outcomes Assessor
Masking Description: An independent adjudication committee (central blinded assessor) will be convened at regular intervals during the study. The adjudication committee will be blinded to study treatment and will review the clinical response assessments at each visit. In case of a discrepancy with the Investigator's assignment of clinical response, the adjudication committee's assessment will prevail.
  In addition, for cIAI subjects classified as a clinical failure, and all cIAI subjects classified as a cure who undergo another procedure (eg, another surgical procedure) subsequent to randomization, the expert panel will review the adequacy of the surgical source control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aztreonam-Avibactam ± Metronidazole (Experimental): All patients randomised to this arm will receive ATM-AVI; all patients with cIAI will receive MTZ for anaerobic cover
  Interventions: Drug: ATM-AVI; Drug: MTZ
- Meropenem ± Colistin (Active Comparator): All patients randomised to this arm will receive MER; addition of COL will be at investigator's discretion in line with local practice
  Interventions: Drug: MER; Drug: COL

INTERVENTIONS:
Drug: ATM-AVI — (Creatinine clearance > 50 mL/min) 6500 mg ATM/2167 mg (loading dose, extended loading dose and maintenance dose) by iv infusion on Day 1 followed by a total daily dose of 6000 mg ATM/2000 mg AVI
  (Creatinine clearance 31 - 50 mL/min) 4250 mg ATM/1417 mg AVI on Day 1 (loading dose, extended loading dose, maintenance dose) followed by total daily dose 3000 mg ATM/1000 mg AVI
  (Creatinine clearance 16 - 30 mL/min) 2700 mg ATM/900 mg AVI on Day 1 (loading dose, extended loading dose maintenance dose), followed by total daily dose 2025 mg ATM/675 mg AVI
  Arms: Aztreonam-Avibactam ± Metronidazole
Drug: MTZ — For cIAI only; 500 mg/100 mL metronidazole iv infusion over 1hr q8h
  Arms: Aztreonam-Avibactam ± Metronidazole
Drug: MER — Where pathogen initially not suspected of being MER-resistant:
  (Creatinine clearance > 50 mL/min) 1000 mg meropenem by 30 min iv infusion q8h
  (Creatinine clearance 26 - 50 mL/min) 1000mg meropenem by 30 min iv infusion q12h
  (Creatinine clearance 16 - 25 mL/min) 500 mg meropenem by 30 min iv infusion q12h
  Where pathogen initially suspected of being MER-resistant (Creatinine clearance > 50 mL/min) 2000 mg meropenem by 180 min iv infusion q8h
  (Creatinine clearance 26 - 50 mL/min) 2000 mg meropenem by 180 min iv infusion q12h
  (Creatinine clearance 16 - 25 mL/min) 1000 mg meropenem by 180 min iv infusion q12h
  Arms: Meropenem ± Colistin
Drug: COL — Loading dose 9 million IU by 30 -60 min iv infusion (6 million IU where weight < 60 kg) followed by one of the following maintenance doses:
  (Creatinine clearance > 50 mL/min) after a 12h interval, commence maintenance dosing 9 million IU daily in 2 or 3 divided doses by 30 -60 min iv infusions.
  (Creatinine clearance 31 - 50 mL/min) After a 24 hr interval, commence maintenance dosing of 6 million IU daily in 2 divided doses by 30 -60 min iv infusion
  (Creatinine clearance 21 - 30 mL/min) After a 24 hr interval, commence maintenance dosing 5 million IU daily in 2 divided doses by 30 -60 min iv infusion
  (Creatinine clearance 16 - 20 mL/min) after a 24 hr interval, commence maintenance dosing 4 million IU daily in 2 divided doses by 30 -60 min iv infusion
  Arms: Meropenem ± Colistin

SUMMARY:
A Phase 3 comparative study to determine the efficacy, safety and tolerability of Aztreonam-Avibactam (ATM-AVI) ± Metronidazole (MTZ) versus Meropenem (MER) ± Colistin (COL) for the treatment of serious infections due to Gram negative bacteria.

DETAILED DESCRIPTION:
A Phase 3 Prospective, Randomized, Multicenter, Open Label, Central Assessor Blinded, Parallel Group, Comparative Study To Determine The Efficacy, Safety And Tolerability Of Aztreonam-Avibactam (ATM-AVI) ± Metronidazole (MTZ) Versus Meropenem±Colistin (MER±COL) For The Treatment Of Serious Infections Due To Gram Negative Bacteria, Including Metallo Β Lactamase (MBL) - Producing Multidrug Resistant Pathogens, For Which There Are Limited Or No Treatment Options

ELIGIBILITY:
Inclusion Criteria:

All subjects:

1. Male or female from 18 years of age
2. Provision of informed consent
3. Confirmed diagnosis of HAP/VAP or cIAI requiring iv antibiotic treatment
4. Female patients are authorized to participate in this clinical study if criteria concerning pregnancy avoidance stated in the protocol are met and negative pregnancy test

Additional for cIAI:

1. Diagnosis of cIAI, EITHER:

   Intra-operative/postoperative enrolment with visual confirmation of cIAI. OR Preoperative enrollment with evidence of systemic inflammatory response, physical and radiological findings consistent with cIAI; confirmation of cIAI at time of surgery within 24 hours of study entry
2. Surgical intervention within 24 hours (before or after) the administration of the first dose of study drug

Additional for HAP/VAP:

1. Onset symptoms > 48h after admission to or <7 days after discharge from an inpatient care facility
2. New or worsening infiltrate on CXR or CT scan
3. Clinical signs and symptoms and laboratory findings consistent with HAP/VAP
4. Respiratory specimen obtained for Gram stain and culture following onset of symptoms and prior to randomisation

Exclusion criteria:

All subjects:

1. APACHE II score > 30
2. Confirmed or suspected infection caused by Gram-negative species not expected to respond to study drug, or Gram-positive species
3. Receipt of >24 hr systemic antibiotic within 48h prior to randomisation (exception in case of treatment failure)
4. History of serious allergy, hypersensitivity (eg, anaphylaxis), or any serious reaction to aztreonam, carbapenem,monobactam or other β-lactam antibiotics, avibactam, nitroimidazoles or metronidazole, or any of the excipients of the study drugs
5. Known Clostridium difficle associated diarrhoea
6. Requirement for effective concomitant systemic antibacterials or antifungals
7. Creatinine clearance ≤15 ml/min or requirement or expectation for renal replacement therapy
8. Acute hepatitis, cirrhosis, acute hepatic failure, chronic hepatic failure
9. Hepatic disease as indicated by AST or ALT >3 × ULN. Patients with AST and/or ALT up to 5 × ULN are eligible if acute and documented by the investigator as being directly related infectious process
10. Patient has a total bilirubin >2 × ULN, unless isolated hyperbilirubinemia is directly related to infectious process or due to known Gilbert's disease
11. ALP >3 × ULN. Patients with values >3 × ULN and <5 x ULN are eligible if acute and directly related to the infectious process being treated
12. Absolute neutrophil count <500/mm3
13. Pregnant or breastfeeding or if of child bearing potential, not using a medically accepted effective method of birth control.
14. Any other condition that may confound the results of the study or pose additional risks to the subject
15. Unlikely to comply with protocol
16. History of epilepsy or seizure disorders excluding febrile seizures of childhood

Additional for cIAI

1. Diagnosis of abdominal wall abscess; small bowel obstruction or ischemic bowel disease without perforation; traumatic bowel perforation with surgery within 12 hours of diagnosis; perforation of gastroduodenal ulcer with surgery < 24 hours of diagnosis primary etiology is not likely to be infectious
2. Simple cholecystitis, gangrenous cholecystitis without rupture, simple appendicitis, acute suppurative cholangitis, infected necrotizing pancreatitis, pancreatic abscess
3. Prior liver, pancreas or small-bowel transplant
4. Staged abdominal repair (STAR), open abdomen technique or marsupialisation

Additional for HAP/VAP

1. APACHE II score < 10
2. Known or high likelihood of Gram-positive monomicrobial infection
3. Lung abscess, pleural empyema, post-obstructive pneumonia
4. Lung or heart transplant
5. Myasthenia gravis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (157):
- United States (5):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
- Argentina (3):
  - Sanatorio Britanico, Rosario, Santa Fe Province
  - Sanatorio Servicios Medicos SM, Santo Tomé, Santa Fe Province
  - Hospital San Roque, Córdoba
- Bulgaria (3):
  - University Hospital Alexandrovska, Clinic of Anesthesiology and Intensive Care, Sofia
  - University Hospital Queen Joanna ISUL, Clinic of Surgery, Sofia
  - University Multiprofile Hospital for Active Treatment ''Prof.Dr Stoyan Kirkovich''AD, Stara Zagora
- China (22):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - The Second People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Nanning First People's Hospital, Nanning, Guangxi
  - Changsha Third Hospital, Changsha, Hunan
  - Hunan Province People's Hospital, Changsha, Hunan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Jiangyin People's Hospital, Jiangyin, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - The First people's Hospital of Kunming, Kunming, Yunnan
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang
  - Quzhou People's Hospital, Quzhou, Zhejiang
  - Peking University People's Hospital, Beijing
  - Jiangyin People's Hospital, Jiangyin
  - Tianjin Union Medical Center, Tianjin
- Croatia (5):
  - Klinicka bolnica Merkur, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Rijeka, Rijeka, Primorje-Gorski Kotar County
  - University Hospital Centre Osijek, Osijek
  - General Hospital "Dr. Josip Bencevic" Slavonski Brod, Slavonski Brod
  - Clinical Hospital Dubrava, Zagreb
- Czechia (6):
  - Fakultni nemocnice Brno, Brno
  - Krajska zdravotni, a.s. - Nemocnice Decin, o.z., Děčín
  - Lekarna Nemocnice Decin, Krajska zdravotni, a.s.- Nemocnice Decin, o.z., Děčín
  - Public Hospital Kolin, a.s., Kolin III
  - Nemocnice Kyjov, prispevkova organizace, Kyjov
  - Fakultni nemocnice Kralovske Vinohrady, Prague
- Greece (7):
  - General Hospital of Athens "Evangelismos", Athens
  - General and Chest Diseases Hospital "Sotiria", Athens
  - General Hospital of Athens "Laiko", Athens
  - University General Hospital "ATTIKON", Athens
  - University General Hospital of Heraklion, Heraklion, Crete
  - University General Hospital of Larissa, Larissa
  - Koutlimbaneio and Triantafylleio General Hospital of Larissa, Larissa
- India (16):
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Victoria Hospital, Bangalore Medical College and Research Institute, Bangalore, Karnataka
  - M S Ramaiah Medical College and Hospitals, Bangalore, Karnataka
  - Kasturba Medical College and Hospital, Manipal, Karnataka
  - JSS Hospital, Mysuru, Karnataka
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Government Medical College, Kozhikode, Kozhikode, Kerala
  - Deenanath Mangeshkar Hospital And Research Centre, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Sahyadri Super Specialty Hospital, Pune, Maharashtra
  - S.R. Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Apollo Hospitals, Chennai, Tamil Nadu
  - King George's Medical University, Lucknow, Uttar Pradesh
  - Dayanand Medical College and Hospital, Ludhiana
  - Sahyadri Clinical Research & Development Center, Pune
  - Sahyadri Specialty Hospital, Pune
- Israel (7):
  - Assuta Ashdod University Hospital, Ashdod
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Organization, Hadassah Medical Center, Ein-Karem, Jerusalem
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
  - Shamir Medical Center, Infectious Diseases Unit, Ẕerifin
- Italy (9):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan, Milan
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti, Foggia
  - Azienda Ospedaliero Universitaria di Modena, Modena
  - Farmacia Ospedaliera - Direzione Assistenza Farmaceutica, Modena
  - SC di Radiologia - Azienda Ospedaliera Universitaria di Modena, Modena
  - Azienda Ospedaliero-Universitaria Pisana Ospedale Cisanello, Pisa
  - UO Radiognastostica 2 Azienda Ospedaliero-Universitaria Pisana Ospedale Cisanello, Pisa
  - UO Farmaceutica Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Azienda Sanitaria Universitaria Friuli Centrale (ASU FC), Presidio Ospedaliero Universitario Santa, Udine
- Malaysia (3):
  - Hospital Seberang Jaya, Seberang Jaya, Pulau Pinang
  - Hospital Sultanah Nur Zahirah, Kuala Terengganu, Terengganu
  - University Malaya Medical Centre, Kuala Lumpur
- Mexico (2):
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
- Philippines (10):
  - De La Salle Medical and Health Sciences Institute, City of Dasmarinas, Cavite
  - Baguio General Hospital and Medical Center, Baguio City
  - Asian Hospital and Medical Center, City of Muntinlupa
  - Davao Doctors Hospital, Davao City
  - St. Paul's Hospital of Iloilo, Inc., Iloilo City
  - West Visayas State University Medical Center, Iloilo City
  - Makati Medical Center, Makati City
  - Philippine General Hospital, Central Intensive Care Unit, Manila
  - Quirino Memorial Medical Center, Quezon City
  - St. Luke's Medical Center, Quezon City
- Romania (5):
  - Institutul National de Boli Infectioase "Prof. Dr. Matei Bals", Bucharest
  - Spitalul Clinic de Boli Infectioase si tropicale "Dr. Victor Babes", Bucharest
  - Spitalul Clinic de Boli Infectioase Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic de Boli Infectioase "Sf. Parascheva" Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta "Pius Brinzeu", Timișoara
- Russia (8):
  - Private Healthcare Institution "Clinical Hospital 'Russian Railroad Medicine, Chelyabinsk'", Chelyabinsk
  - State Budgetary Healthcare Institution "Regional Clinical Hospital No. 2" of the Ministry of Health, Krasnodar
  - GBUZ of Novosibirsk region "City Clinical Hospital # 2", Novosibirsk
  - State autonomous institution of healthcare of the Perm Region" City clinical hospital #4", Perm
  - FGBOU VO "The First St. Petersburg state medical university n. a. I.P. Pavlova", Saint Petersburg
  - OGBUZ "Smolensk Regional Clinical Hospital", Smolensk
  - FSBEI of HE "Smolensk State Medical University" of the Ministry of Health of the RF, Smolensk
  - Scientific Research Institute of Antimicrobial Chemotherapy, Smolensk
- South Korea (4):
  - Gachon University Gil Medical Center - Infectious Disease, Incheon, Incheon Gwang'yeogsiv
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
- Spain (12):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Mutua de Terrassa, Terrassa, Barcelona
  - Complejo Hospitalario Universitario de Vigo. Area Sanitaria de Vigo. Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Parc de Salut Mar- Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic la Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (6):
  - National Taiwan University Hospital Yun-Lin Branch, Douliu, Yunlin
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
- Thailand (4):
  - Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok
  - Srinagarind Hospital, Division of Infectious Disease and Tropical Medicine, Muang, Changwat Khon Kaen
  - Bamrasnaradura Infectious Disease Institute (BIDI), Muang, Changwat Nonthaburi
  - Songklanagarind Hospital, Prince of Songkla University, Hat Yai, Changwat Songkhla
- Turkey (Türkiye) (8):
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Ankara University Faculty of Medicine, Ankara
  - T.C. Saglik Bakanligi Ankara Sehir Hastanesi, Ankara
  - Acibadem Atakent Hospital, Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi, Istanbul
  - Ege University Faculty of Medicine, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Karadeniz Technical University Medical Faculty Farabi Hospital, Trabzon
- Ukraine (12):
  - OKU "Chernivetska oblasna klinichna likarnia", khirurhichne viddilennia, Chernivtsi
  - KZ "Dnipropetrovska oblasna klinichna likarnia im. I.I. Mechnykova", viddilennia khirurhii №2, Dnipro
  - Komunalnyi zaklad "Miska klinichna likarnia No.4" Dniprovskoi miskoi rady, viddilennia profpatolohii, Dnipro
  - Oblasna klinichna likarnia, viddilennia anesteziolohii ta intensyvnoi terapii, Ivano-Frankivsk
  - Ivano-Frankivska tsentralna miska klin likarnia, viddilennia khirurhii,, Ivano-Frankivsk
  - DU "Instytut zahalnoi ta nevidkladnoi khirurhii imeni V.T. Zaitseva Natsionalnoi akademii medychnykh, Kharkiv
  - Kyivska miska klinichna likarnia No. 3, khirurhichne viddilennia, Kyiv
  - Kyivska miska klinichna likarnia #4, khirurhichne viddilennia #1, Kyiv
  - Komunalne nekomertsiine pidpryiemstvo Lvivskoi oblasnoi rady Lvivska oblasna klinichna likarnia, Lviv
  - Odeska klinichna likarnia na zaliznychnomu transporti filii "Tsentr okhorony zdorovia" aktsionernoho, Odesa
  - Komunalne pidpryiemstvo "1-a miska klinichna likarnia Poltavskoi miskoi rady",, Poltava
  - Vinnytska oblasna klinichna likarnia im. M.I. Pyrohova, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Raber SR, Xie R, Rogers H, Soto E, Arhin FF, Stone GG, Leister-Tebbe H, Chow JW. Microbiological, Clinical, and Pharmacokinetic/Pharmacodynamic Data to Support EUCAST Aztreonam-Avibactam Minimum Inhibitory Concentration Susceptibility Breakpoints Against Enterobacterales. Infect Dis Ther. 2026 Jan;15(1):183-195. doi: 10.1007/s40121-025-01267-3. Epub 2025 Nov 21. PMID 41269522
- [Derived] Xie R, Rogers H, Chow JW, Soto E, Raber SR. Population pharmacokinetic/pharmacodynamic modeling to optimize aztreonam-avibactam dose regimens for adult patients. Antimicrob Agents Chemother. 2025 Aug 6;69(8):e0195024. doi: 10.1128/aac.01950-24. Epub 2025 Jun 18. PMID 40530972
- [Derived] Carmeli Y, Cisneros JM, Paul M, Daikos GL, Wang M, Torre-Cisneros J, Singer G, Titov I, Gumenchuk I, Zhao Y, Jimenez-Rodriguez RM, Liang L, Chen G, Pyptiuk O, Aksoy F, Rogers H, Wible M, Arhin FF, Luckey A, Leaney JL, Pypstra R, Chow JW; COMBACTE-CARE consortium REVISIT study group. Aztreonam-avibactam versus meropenem for the treatment of serious infections caused by Gram-negative bacteria (REVISIT): a descriptive, multinational, open-label, phase 3, randomised trial. Lancet Infect Dis. 2025 Feb;25(2):218-230. doi: 10.1016/S1473-3099(24)00499-7. Epub 2024 Oct 7. PMID 39389071
- [Derived] Das S, Riccobene T, Carrothers TJ, Wright JG, MacPherson M, Cristinacce A, McFadyen L, Xie R, Luckey A, Raber S. Dose selection for aztreonam-avibactam, including adjustments for renal impairment, for Phase IIa and Phase III evaluation. Eur J Clin Pharmacol. 2024 Apr;80(4):529-543. doi: 10.1007/s00228-023-03609-x. Epub 2024 Jan 22. PMID 38252170
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3601002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were hospitalized with a diagnosis of complicated intra-abdominal infection (cIAI) or nosocomial pneumonia (NP) including hospital-acquired pneumonia (HAP) and ventilator-associated pneumonia (VAP) were enrolled. This study was conducted across 20 countries from 05-Apr-2018 to 23-Feb-2023.
Pre-assignment Details: A total of 461 participants were screened of which 38 failed screening and 1 participant was not randomized due to lack of study drug at the site. A total of 422 participants were randomized in the study.
Groups:
- Aztreonam-avibactam ± Metronidazole: Participants hospitalized with cIAI or NP (including HAP and VAP) were randomized to receive a loading dose of aztreonam-avibactam (ATM-AVI) by intravenous (IV) infusion over 30 minutes, immediately followed by an extended loading dose of ATM-AVI by IV infusion over 3 hours on Day 1. Participants were administered a maintenance dose of ATM-AVI by IV infusion over 3 hours on Days 2 to 14. Participants with cIAI also received metronidazole (MTZ) 500 milligrams (mg) IV every 8 hours.
- Meropenem± Colistimethate: Participants hospitalized with cIAI or NP (including HAP and VAP) were randomized to receive 1000 mg meropenem every 8 hours by IV infusion. A higher dose of 2000 mg was given by IV infusion over 180 minutes if carbapenem resistant pathogen was strongly suspected. Participants were administered colistimethate sodium at investigator's discretion.
Period: Overall Study
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Started | 282 | 140
Participants With cIAI | 208 | 104
Participants With HAP/VAP | 74 | 36
Completed | 242 | 122
Not Completed | 40 | 18
Not completed — Other | 2 | 2
Not completed — Withdrawal by Subject | 16 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Death | 17 | 11
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) analysis set included all randomized participants regardless of receipt of study drug. Participants were analyzed according to the treatment to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate | Total
Number analyzed (Participants) | 282 | 140 | 422
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.2 (17.84) | 54.0 (16.30) | 54.8 (17.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 39 | 135
  Male | 186 | 101 | 287
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58 | 21 | 79
  Not Hispanic or Latino | 213 | 113 | 326
  Unknown or Not Reported | 11 | 6 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 164 | 64 | 228
  Black or African American | 1 | 1 | 2
  Asian | 107 | 69 | 176
  American Indian or Alaska Native | 7 | 2 | 9
  Mixed | 2 | 1 | 3
  Other | 0 | 1 | 1
  Not reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Cure at Test of Cure (TOC) Visit: Intent-To-Treat (ITT) Analysis Set
Description: Clinical cure was defined as improvement in baseline signs and symptoms such that after study treatment, no further antimicrobial treatment for the index infection (i.e., cIAI or HAP/VAP) was required. Additionally, for cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. Clinical cure was determined by the Independent Clinical Adjudication Committee. 95% confidence interval (CI) was based on Jeffrey's method.
Time Frame: At TOC visit (Day 28)
Population: The ITT analysis set included all randomized participants regardless of receipt of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 282 | 140
Percentage of participants | 68.4 [62.8 to 73.7] | 65.7 [57.6 to 73.2]
Statistical Analysis 1: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; Test type: Other; Difference in clinical cure rate = 2.7, 95% CI 2-sided [-6.6 to 12.4] — The confidence interval (CI) for the difference was calculated using the unstratified Miettinen and Nurminen method

2. Primary Outcome: Percentage of Participants With Clinical Cure at TOC Visit: Clinically Evaluable (CE) Analysis Set
Description: Clinical cure = improvement in baseline signs and symptoms such that after study treatment, no further antimicrobial treatment for the index infection (i.e., cIAI or HAP/VAP) was required. Additionally for cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. Clinical cure was determined by Independent Clinical Adjudication Committee. 95% CI was based on Jeffrey's method. CE analysis set:all participants in ITT analysis set; met criteria for cIAI, or HAP/VAP; received at least 48 hours of study treatment or <48 hours of treatment before discontinuing study drug due to AE; no concomitant antibiotics for any baseline pathogens between first dose and TOC (except protocol-allowed antibiotics); no prior antibiotics other than allowed per protocol; no important protocol deviations; no clinical outcome of indeterminate at TOC; no monomicrobial infections due to non-eligible pathogens and did not have only Gram-positive pathogens.
Time Frame: At TOC visit (Day 28)
Population: Analysis was performed on CE analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 213 | 105
Percentage of participants | 77.0 [71.0 to 82.3] | 74.3 [65.3 to 81.9]
Statistical Analysis 1: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; Test type: Other; Difference in clinical cure rate = 2.7, 95% CI 2-sided [-7.0 to 13.2] — The CI for the difference was calculated using the unstratified Miettinen and Nurminen method

3. Secondary Outcome: Percentage of Participants With Clinical Cure at TOC Visit: Microbiological Intent-To-Treat (Micro-ITT) Analysis Set
Description: Clinical cure was defined as improvement in baseline signs and symptoms such that after study treatment, no further antimicrobial treatment for the index infection (i.e., cIAI or HAP/VAP) was required. Additionally, for cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. Clinical cure was determined by the Independent Clinical Adjudication Committee. 95% CI was based on Jeffrey's method.
Time Frame: At TOC visit (Day 28)
Population: The microbiological Intent-To-Treat (micro-ITT) analysis set was a subset of the ITT analysis set and included all participants who had at least one Gram-negative baseline pathogen from an adequate specimen obtained prior to the start of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 177 | 94
Percentage of participants | 72.9 [66.0 to 79.0] | 72.3 [62.7 to 80.6]
Statistical Analysis 1: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; Test type: Other; Difference in clinical cure rate = 0.5, 95% CI 2-sided [-10.2 to 12.1] — CI for the difference was calculated using the unstratified Miettinen and Nurminen method

4. Secondary Outcome: Percentage of Participants With Clinical Cure at TOC Visit: Microbiologically Evaluable (ME) Analysis Set
Description: as for outcome 3
Time Frame: At TOC visit (Day 28)
Population: ME analysis set included all participants commonly included in both micro-ITT and CE analysis sets and included participants who had at least 1 etiologic pathogen from an adequate baseline culture regardless of susceptibility to study agents.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 149 | 79
Percentage of participants | 78.5 [71.4 to 84.5] | 75.9 [65.7 to 84.3]
Statistical Analysis 1: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; Test type: Other; Difference in clinical cure rate = 2.6, 95% CI 2-sided [-8.4 to 14.7] — CI for the difference was calculated using the unstratified Miettinen and Nurminen method

5. Secondary Outcome: Percentage of Participants With Clinical Cure at TOC Visit by Type of Infection: ITT Analysis Set
Description: as for outcome 3
Time Frame: At TOC visit (Day 28)
Population: ITT analysis set included all randomized participants regardless of receipt of study drug. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 282 | 140
Percentage of participants
  cIAI: number analyzed (Participants) | 208 | 104
  cIAI | 76.4 [70.3 to 81.8] | 74.0 [65.0 to 81.7]
  HAP/VAP: number analyzed (Participants) | 74 | 36
  HAP/VAP | 45.9 [34.9 to 57.3] | 41.7 [26.7 to 57.9]
Statistical Analysis 1: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; cIAI; Test type: Other; Difference in clinical cure rate = 2.4, 95% CI 2-sided [-7.4 to 13.0] — CI for the difference was calculated using the unstratified Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; HAP/VAP; Test type: Other; Difference; Difference in clinical cure rate = 4.3, 95% CI 2-sided [-15.5 to 23.1] — CI for the difference was calculated using the unstratified Miettinen and Nurminen method

6. Secondary Outcome: Percentage of Participants With Clinical Cure at TOC Visit by Type of Infection: CE Analysis Set
Description: Clinical cure = improvement in baseline signs and symptoms such that after study treatment, no further antimicrobial treatment for the index infection (i.e., cIAI or HAP/VAP) was required. Additionally, for cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. Clinical cure was determined by the Independent Clinical Adjudication Committee. 95% CI was based on Jeffrey's method. CE analysis set:all participants in ITT analysis set; met criteria for cIAI, or HAP/VAP; received at least 48 hours of study treatment or <48 hours of treatment before discontinuing study drug due to AE; no concomitant antibiotics for any baseline pathogens between first dose and TOC (except protocol-allowed antibiotics); no prior antibiotics other than allowed per protocol; no important protocol deviations; no clinical outcome of indeterminate at TOC; no monomicrobial infections due to non-eligible pathogens and did not have only Gram-positive pathogens.
Time Frame: At TOC visit (Day 28)
Population: CE analysis set. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 213 | 105
Percentage of participants
  cIAI: number analyzed (Participants) | 168 | 83
  cIAI | 85.1 [79.2 to 89.9] | 79.5 [69.9 to 87.1]
  HAP/VAP: number analyzed (Participants) | 45 | 22
  HAP/VAP | 46.7 [32.7 to 61.1] | 54.5 [34.3 to 73.7]
Statistical Analysis 1: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; cIAI; Test type: Other; Difference in clinical cure rate = 5.6, 95% CI 2-sided [-4.0 to 16.6] — CI for the difference was calculated using the unstratified Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; HAP/VAP; Test type: Other; Difference in clinical cure rate = -7.9, 95% CI 2-sided [-31.9 to 17.3] — CI for the difference was calculated using the unstratified Miettinen and Nurminen method

7. Secondary Outcome: Percentage of Participants With Clinical Cure in Participants With Metallo-beta-lactamase (MBL) Positive Pathogen at TOC Visit: Micro-ITT Analysis Set
Description: Clinical cure was defined as improvement in baseline signs and symptoms such that after study treatment, no further antimicrobial treatment for the index infection (i.e., cIAI or HAP/VAP) was required. Additionally, for cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. Clinical cure was determined by the Independent Clinical Adjudication Committee.
Time Frame: At TOC visit (Day 28)
Population: Micro-ITT analysis set was a subset of the ITT analysis and included all participants who had at least 1 Gram-negative baseline pathogen from an adequate specimen obtained prior to the start of study treatment. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 7 | 3
Percentage of participants | 28.6 | 66.7

8. Secondary Outcome: Percentage of Participants With Clinical Cure in Participants With MBL Positive Pathogen at TOC Visit: ME Analysis Set
Description: Clinical cure was defined as improvement in baseline signs and symptoms such that after study treatment, no further antimicrobial treatment for the index infection (i.e., cIAI or HAP/VAP) was required. For cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. Clinical cure was determined by the Independent Clinical Adjudication Committee.
Time Frame: At TOC visit (Day 28)
Population: The ME analysis set included all participants commonly included in both micro-ITT and CE analysis sets and included participants who had at least 1 etiologic pathogen from an adequate baseline culture regardless of susceptibility to study agents. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 4 | 1
Percentage of participants | 50.0 | 0

9. Secondary Outcome: Percentage of Participants With Favorable Per-Participant Microbiological Response at TOC Visit: Micro- ITT Analysis Set
Description: Participants were determined to have a favorable microbiological response if all baseline pathogens for that participant had a favorable outcome (eradicated or presumed eradicated). Eradication: Absence of causative pathogen from an appropriately obtained specimen at the site of infection. Presumed eradication: repeat culture of specimens were not performed/clinically indicated in a participant who had a clinical response of cure.
Time Frame: At TOC visit day (28)
Population: Micro-ITT analysis set was a subset of the ITT analysis sets and included all participants who had at least 1 Gram-negative baseline pathogen from an adequate specimen obtained prior to the start of study treatment. Participants with a per participant response of indeterminate were excluded from this analysis. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 169 | 92
Percentage of participants | 75.7 | 73.9

10. Secondary Outcome: Percentage of Participants With Favorable Per-Participant Microbiological Response at TOC Visit: ME Analysis Set
Description: as for outcome 9
Time Frame: At TOC Visit (Day 28)
Population: The ME analysis set included all participants commonly included in both micro-ITT and CE analysis sets and included participants who had at least 1 etiologic pathogen from an adequate baseline culture regardless of susceptibility to study agents.
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 149 | 79
Percentage of participants | 77.2 | 75.9

11. Secondary Outcome: Percentage of Participants Who Died on or Before 28 Days After Randomization: ITT Analysis Set
Description: Percentage of participants who died on or before 28 days after randomization is reported in this outcome measure.
Time Frame: From randomization up to 28 days
Population: The ITT analysis set included all randomized participants regardless of receipt of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 282 | 140
Percentage of participants | 4.3 | 7.1

12. Secondary Outcome: Percentage of Participants Who Died on or Before 28 Days After Randomization: Micro-ITT Analysis Set
Description: Percentage of participants who died on or before 28 days after randomization is reported in this outcome measure.
Time Frame: From randomization up to 28 days
Population: Micro-ITT analysis set was a subset of the ITT analysis set and included all participants who had at least 1 Gram-negative baseline pathogen from an adequate specimen obtained prior to the start of study treatment.
Measure: Number; unit: Percenatge of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 177 | 94
Percenatge of participants | 2.8 | 6.4

13. Secondary Outcome: Plasma Concentration of Aztreonam
Description: Plasma concentration for aztreonam according to renal function (augmented, normal and mild, moderate and severe is presented in this outcome measure. Augmented = Creatinine clearance (CrCL) > 150 milliliters per minute (mL/min); Normal & Mild = CrCL > 50 to <=150 mL/min; Moderate = CrCL > 30 to ≤ 50 mL/min; Severe = CrCL > 15 to ≤ 30 mL/min.
Time Frame: Anytime between 25 to 30 minutes, 3.25 to 3.5 hours, 5.5 to 6.5 hours, 7.5 to 8.5 hours post start of infusion on Day 1; 2.75 to 3 hours, 3.5 to 4.5 hours, 5 to 6 and 7 to 8 hours post start of infusion on Day 4
Population: PK analysis set included all participants who had at least 1 plasma concentration data assessment available for ATM or AVI. All participants reported under 'Overall Number of Participants Analyzed' included participants evaluable for this outcome measure and contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligram/Liter
Arm/Group | Aztreonam-avibactam ± Metronidazole
Number analyzed (Participants) | 253
Milligram/Liter
  Renal Function: Augmented:25 to 30 minutes post start of infusion on Day 1: number analyzed (Participants) | 36
  Renal Function: Augmented:25 to 30 minutes post start of infusion on Day 1 | 43.3 (339.08)
  Renal Function: Augmented:3.25 to 3.5 hours post start of infusion on Day 1: number analyzed (Participants) | 34
  Renal Function: Augmented:3.25 to 3.5 hours post start of infusion on Day 1 | 55.99 (287.36)
  Renal Function: Augmented: 5.5 hours to 6.5 hours post loading infusion on Day 1: number analyzed (Participants) | 34
  Renal Function: Augmented: 5.5 hours to 6.5 hours post loading infusion on Day 1 | 26.11 (338.5)
  Renal Function: Augmented: 7.5 to 8.5 hours post start of infusion on Day 1: number analyzed (Participants) | 0
  Renal Function: Normal & Mild: 25 to 30 min post start of infusion on Day 1: number analyzed (Participants) | 169
  Renal Function: Normal & Mild: 25 to 30 min post start of infusion on Day 1 | 33.85 (234.46)
  Renal Function: Normal & Mild:3.25 to 3.5 hours post start of infusion on Day 1: number analyzed (Participants) | 164
  Renal Function: Normal & Mild:3.25 to 3.5 hours post start of infusion on Day 1 | 56.24 (222.32)
  Renal Function: Normal & Mild:5.5 hours to 6.5 hours post start of infusion on Day 1: number analyzed (Participants) | 160
  Renal Function: Normal & Mild:5.5 hours to 6.5 hours post start of infusion on Day 1 | 25.03 (115.83)
  Renal Function: Normal & Mild:7.5 to 8.5 hours post start of infusion on Day 1: number analyzed (Participants) | 7
  Renal Function: Normal & Mild:7.5 to 8.5 hours post start of infusion on Day 1 | 34.62 (54.42)
  Renal Function: Moderate: 25 to 30 min post start of infusion on Day 1: number analyzed (Participants) | 25
  Renal Function: Moderate: 25 to 30 min post start of infusion on Day 1 | 54.49 (313.99)
  Renal Function: Moderate: 3.25 to 3.5 hours post start of infusion on Day 1: number analyzed (Participants) | 24
  Renal Function: Moderate: 3.25 to 3.5 hours post start of infusion on Day 1 | 73.72 (259.64)
  Renal Function: Moderate: 5.5 hours to 6.5 hours post start of infusion on Day 1: number analyzed (Participants) | 20
  Renal Function: Moderate: 5.5 hours to 6.5 hours post start of infusion on Day 1 | 52.45 (139.9)
  Renal Function: Moderate: 7.5 to 8.5 hours post start of infusion on Day 1: number analyzed (Participants) | 1
  Renal Function: Moderate: 7.5 to 8.5 hours post start of infusion on Day 1 | 34 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed.
  Renal Function: Severe: 25 to 30 min post start of infusion on Day 1: number analyzed (Participants) | 8
  Renal Function: Severe: 25 to 30 min post start of infusion on Day 1 | 48.98 (187.86)
  Renal Function: Severe: 3.25 to 3.5 hours post start of infusion on Day 1: number analyzed (Participants) | 8
  Renal Function: Severe: 3.25 to 3.5 hours post start of infusion on Day 1 | 50.31 (30.13)
  Renal Function: Severe: 5.5 hours to 6.5 hours post start of infusion on Day 1: number analyzed (Participants) | 2
  Renal Function: Severe: 5.5 hours to 6.5 hours post start of infusion on Day 1 | 48.54 (46.87)
  Renal Function: Severe: 7.5 to 8.5 hours post start of infusion on Day 1: number analyzed (Participants) | 5
  Renal Function: Severe: 7.5 to 8.5 hours post start of infusion on Day 1 | 29.42 (34.88)
  Renal Function: Augmented: 2.75 to 3 hours post start of infusion on Day 4: number analyzed (Participants) | 33
  Renal Function: Augmented: 2.75 to 3 hours post start of infusion on Day 4 | 46.11 (234.31)
  Renal Function: Augmented: 3.5 to 4.5 hours post start of infusion on Day 4: number analyzed (Participants) | 38
  Renal Function: Augmented: 3.5 to 4.5 hours post start of infusion on Day 4 | 33.56 (204.99)
  Renal Function: Augmented: 5 to 6 hours post start of infusion on Day 4: number analyzed (Participants) | 38
  Renal Function: Augmented: 5 to 6 hours post start of infusion on Day 4 | 19.56 (205.84)
  Renal Function: Augmented: 7 to 8 hours post start of infusion on Day 4: number analyzed (Participants) | 1
  Renal Function: Augmented: 7 to 8 hours post start of infusion on Day 4 | 14.1 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed.
  Renal Function: Normal & Mild: 2.75 to 3 hours post start of infusion on Day 4: number analyzed (Participants) | 163
  Renal Function: Normal & Mild: 2.75 to 3 hours post start of infusion on Day 4 | 56.59 (404.54)
  Renal Function: Normal & Mild: 3.5 to 4.5 hours post start of infusion on Day 4: number analyzed (Participants) | 168
  Renal Function: Normal & Mild: 3.5 to 4.5 hours post start of infusion on Day 4 | 35.69 (422.52)
  Renal Function: Normal & Mild: 5 to 6 hours post start of infusion on Day 4: number analyzed (Participants) | 154
  Renal Function: Normal & Mild: 5 to 6 hours post start of infusion on Day 4 | 21.75 (271.62)
  Renal Function: Normal & Mild: 7 to 8 hours post start of infusion on Day 4: number analyzed (Participants) | 6
  Renal Function: Normal & Mild: 7 to 8 hours post start of infusion on Day 4 | 42.98 (62.54)
  Renal Function: Moderate: 2.75 to 3 hours post start of infusion on Day 4: number analyzed (Participants) | 24
  Renal Function: Moderate: 2.75 to 3 hours post start of infusion on Day 4 | 73.33 (183.2)
  Renal Function: Moderate: 3.5 to 4.5 hours post start of infusion on Day 4: number analyzed (Participants) | 24
  Renal Function: Moderate: 3.5 to 4.5 hours post start of infusion on Day 4 | 58 (129.36)
  Renal Function: Moderate: 5 to 6 hours post start of infusion on Day 4: number analyzed (Participants) | 22
  Renal Function: Moderate: 5 to 6 hours post start of infusion on Day 4 | 44.72 (59.15)
  Renal Function: Moderate: 7 to 8 hours post start of infusion on Day 4: number analyzed (Participants) | 1
  Renal Function: Moderate: 7 to 8 hours post start of infusion on Day 4 | 19.8 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed.
  Renal Function: Severe: 2.75 to 3 hours post start of infusion on Day 4: number analyzed (Participants) | 7
  Renal Function: Severe: 2.75 to 3 hours post start of infusion on Day 4 | 54.91 (45.17)
  Renal Function: Severe: 3.5 to 4.5 hours post start of infusion on Day 4: number analyzed (Participants) | 6
  Renal Function: Severe: 3.5 to 4.5 hours post start of infusion on Day 4 | 45.17 (34.89)
  Renal Function: Severe: 5 to 6 hours post start of infusion on Day 4: number analyzed (Participants) | 4
  Renal Function: Severe: 5 to 6 hours post start of infusion on Day 4 | 45.11 (57.13)
  Renal Function: Severe:7 to 8 hours post start of infusion on Day 4: number analyzed (Participants) | 4
  Renal Function: Severe:7 to 8 hours post start of infusion on Day 4 | 32.69 (55.56)

14. Secondary Outcome: Plasma Concentration of Avibactam
Description: Plasma concentration for avibactam according to renal function (augmented, normal and mild, moderate and severe is presented in this outcome measure. Augmented = CrCL > 150 mL/min; Normal & Mild = CrCL > 50 to <=150 mL/min; Moderate = CrCL > 30 to ≤ 50 mL/min; Severe = CrCL > 15 to ≤ 30 mL/min.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligram/Liter
Arm/Group | Aztreonam-avibactam ± Metronidazole
Number analyzed (Participants) | 235
Milligram/Liter
  Renal Function: Augmented:25 to 30 minutes post start of infusion on Day 1: number analyzed (Participants) | 36
  Renal Function: Augmented:25 to 30 minutes post start of infusion on Day 1 | 10.77 (353.86)
  Renal Function: Augmented:3.25 to 3.5 hours post start of infusion on Day 1: number analyzed (Participants) | 34
  Renal Function: Augmented:3.25 to 3.5 hours post start of infusion on Day 1 | 12.6 (299.27)
  Renal Function: Augmented: 5.5 hours to 6.5 hours post start of infusion on Day 1: number analyzed (Participants) | 34
  Renal Function: Augmented: 5.5 hours to 6.5 hours post start of infusion on Day 1 | 4.75 (366.33)
  Renal Function: Augmented:7.5 to 8.5 hours post start of infusion on Day 1: number analyzed (Participants) | 0
  Renal Function: Normal & Mild: 25 to 30 min post start of infusion on Day 1: number analyzed (Participants) | 170
  Renal Function: Normal & Mild: 25 to 30 min post start of infusion on Day 1 | 8.81 (338.73)
  Renal Function: Normal & Mild:3.25 to 3.5 hours post start of infusion on Day 1: number analyzed (Participants) | 164
  Renal Function: Normal & Mild:3.25 to 3.5 hours post start of infusion on Day 1 | 13.76 (242.67)
  Renal Function: Normal & Mild:5.5 hours to 6.5 hours post start of infusion on Day 1: number analyzed (Participants) | 160
  Renal Function: Normal & Mild:5.5 hours to 6.5 hours post start of infusion on Day 1 | 4.85 (209.49)
  Renal Function: Normal & Mild:7.5 to 8.5 hours post start of infusion on Day 1: number analyzed (Participants) | 7
  Renal Function: Normal & Mild:7.5 to 8.5 hours post start of infusion on Day 1 | 7.18 (62.62)
  Renal Function: Moderate: 25 to 30 min post start of infusion on Day 1: number analyzed (Participants) | 25
  Renal Function: Moderate: 25 to 30 min post start of infusion on Day 1 | 13.56 (383.79)
  Renal Function: Moderate: 3.25 to 3.5 hours post start of infusion on Day 1: number analyzed (Participants) | 24
  Renal Function: Moderate: 3.25 to 3.5 hours post start of infusion on Day 1 | 20.28 (262.6)
  Renal Function: Moderate: 5.5 hours to 6.5 hours post start of infusion on Day 1: number analyzed (Participants) | 20
  Renal Function: Moderate: 5.5 hours to 6.5 hours post start of infusion on Day 1 | 13.47 (160.75)
  Renal Function: Moderate: 7.5 to 8.5 hours post start of infusion on Day 1: number analyzed (Participants) | 1
  Renal Function: Moderate: 7.5 to 8.5 hours post start of infusion on Day 1 | 7.91 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed.
  Renal Function: Severe: 25 to 30 min post start of infusion on Day 1: number analyzed (Participants) | 8
  Renal Function: Severe: 25 to 30 min post start of infusion on Day 1 | 14.11 (202.08)
  Renal Function: Severe: 3.25 to 3.5 hours post start of infusion on Day 1: number analyzed (Participants) | 8
  Renal Function: Severe: 3.25 to 3.5 hours post start of infusion on Day 1 | 13.62 (39.68)
  Renal Function: Severe: 5.5 hours to 6.5 hours post start of infusion on Day 1: number analyzed (Participants) | 2
  Renal Function: Severe: 5.5 hours to 6.5 hours post start of infusion on Day 1 | 11.6 (54.34)
  Renal Function: Severe: 7.5 to 8.5 hours post start of infusion on Day 1: number analyzed (Participants) | 5
  Renal Function: Severe: 7.5 to 8.5 hours post start of infusion on Day 1 | 8 (57.91)
  Renal Function: Augmented: 2.75 to 3 hours post start of infusion on Day 4: number analyzed (Participants) | 33
  Renal Function: Augmented: 2.75 to 3 hours post start of infusion on Day 4 | 9.75 (289.96)
  Renal Function: Augmented: 3.5 to 4.5 hours post start of infusion on Day 4: number analyzed (Participants) | 38
  Renal Function: Augmented: 3.5 to 4.5 hours post start of infusion on Day 4 | 6.23 (263.94)
  Renal Function: Augmented: 5 to 6 hours post start of infusion on Day 4: number analyzed (Participants) | 38
  Renal Function: Augmented: 5 to 6 hours post start of infusion on Day 4 | 3.19 (265.65)
  Renal Function: Augmented: 7 to 8 hours post start of infusion on Day 4: number analyzed (Participants) | 1
  Renal Function: Augmented: 7 to 8 hours post start of infusion on Day 4 | 2.72 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed.
  Renal Function: Normal & Mild: 2.75 to 3 hours post start of infusion on Day 4: number analyzed (Participants) | 163
  Renal Function: Normal & Mild: 2.75 to 3 hours post start of infusion on Day 4 | 11.46 (504.77)
  Renal Function: Normal & Mild: 3.5 to 4.5 hours post start of infusion on Day 4: number analyzed (Participants) | 168
  Renal Function: Normal & Mild: 3.5 to 4.5 hours post start of infusion on Day 4 | 6.29 (493.48)
  Renal Function: Normal & Mild: 5 to 6 hours post start of infusion on Day 4: number analyzed (Participants) | 154
  Renal Function: Normal & Mild: 5 to 6 hours post start of infusion on Day 4 | 3.48 (382.3)
  Renal Function: Normal & Mild: 7 to 8 hours post start of infusion on Day 4: number analyzed (Participants) | 6
  Renal Function: Normal & Mild: 7 to 8 hours post start of infusion on Day 4 | 6.19 (51.22)
  Renal Function: Moderate: 2.75 to 3 hours post start of infusion on Day 4: number analyzed (Participants) | 24
  Renal Function: Moderate: 2.75 to 3 hours post start of infusion on Day 4 | 16.98 (208.63)
  Renal Function: Moderate: 3.5 to 4.5 hours post start of infusion on Day 4: number analyzed (Participants) | 24
  Renal Function: Moderate: 3.5 to 4.5 hours post start of infusion on Day 4 | 12.86 (156.96)
  Renal Function: Moderate: 5 to 6 hours post start of infusion on Day 4: number analyzed (Participants) | 22
  Renal Function: Moderate: 5 to 6 hours post start of infusion on Day 4 | 9.23 (72.89)
  Renal Function: Moderate: 7 to 8 hours post start of infusion on Day 4: number analyzed (Participants) | 1
  Renal Function: Moderate: 7 to 8 hours post start of infusion on Day 4 | 4.35 (NA) — Geometric coefficient of variation could not be estimated as only 1 participant was analyzed.
  Renal Function: Severe: 2.75 to 3 hours post start of infusion on Day 4: number analyzed (Participants) | 7
  Renal Function: Severe: 2.75 to 3 hours post start of infusion on Day 4 | 14.35 (44.72)
  Renal Function: Severe: 3.5 to 4.5 hours post start of infusion on Day 4: number analyzed (Participants) | 6
  Renal Function: Severe: 3.5 to 4.5 hours post start of infusion on Day 4 | 11.68 (42.15)
  Renal Function: Severe: 5 to 6 hours post start of infusion on Day 4: number analyzed (Participants) | 4
  Renal Function: Severe: 5 to 6 hours post start of infusion on Day 4 | 9.99 (67.87)
  Renal Function: Severe: Moderate: 7 to 8 hours post start of infusion on Day 4: number analyzed (Participants) | 4
  Renal Function: Severe: Moderate: 7 to 8 hours post start of infusion on Day 4 | 8.97 (47.28)

15. Secondary Outcome: Maximum Plasma Concentration for a Dosing Interval at Steady-State (Cmax, ss) According to Clinical Response by Infection Type at TOC: Aztreonam
Description: Population PK predicted maximum plasma concentration for a dosing interval at steady-state (Cmax,ss) for participants who received aztreonam-avibactam in studies C3601002 (NCT03329092) and C3601009 (NCT03580044). Clinical response categories included, clinical cure=improvement in baseline signs and symptoms such that after study treatment, no further antimicrobial treatment for the index infection (i.e., cIAI or HAP/VAP) was required. For cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. Failure was defined as participants who met any of the following criteria like death (after receiving at least 48 hours of study treatment) and participants who received treatment with further antibiotics for the index infection. Indeterminate was defined as death (after receiving less than 48 hours of study treatment) and for cIAI participants inadequate infection source control at time of initial surgical procedure.
Time Frame: At TOC (Day 28)
Population: Analysis population included participants from PK and ITT analysis set. All participants reported under 'Overall Number of Participants Analyzed' included participants evaluable for this outcome measure and contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligram per liter (mg/L)
Groups:
- Aztreonam- Avibactam: Participants who received aztreonam-avibactam in studies C3601002 (NCT03329092) and C3601009 (NCT03580044) were included in the analysis.
Arm/Group | Aztreonam- Avibactam
Number analyzed (Participants) | 262
Milligram per liter (mg/L)
  cIAI: Clinical cure: number analyzed (Participants) | 151
  cIAI: Clinical cure | 52.47 (37.49)
  cIAI: Failure: number analyzed (Participants) | 31
  cIAI: Failure | 56.71 (62.52)
  cIAI: Indeterminate: number analyzed (Participants) | 9
  cIAI: Indeterminate | 66.21 (12.7)
  HAP:Clinical cure: number analyzed (Participants) | 17
  HAP:Clinical cure | 85.24 (48.49)
  HAP: Failure: number analyzed (Participants) | 16
  HAP: Failure | 64.57 (33.97)
  HAP: Indeterminate: number analyzed (Participants) | 5
  HAP: Indeterminate | 61.79 (27.2)
  VAP: Clinical Cure: number analyzed (Participants) | 16
  VAP: Clinical Cure | 54.89 (30.42)
  VAP: Failure: number analyzed (Participants) | 16
  VAP: Failure | 56.5 (31.1)
  VAP: Indeterminate: number analyzed (Participants) | 1
  VAP: Indeterminate | 85.34 (NA) — Standard deviation (SD) was not estimated because of less number of participants in this event.

16. Secondary Outcome: Percentage of Time That Free Plasma Concentrations Are Above the Minimum Inhibitory Concentration Over a Dosing Interval (%fT>MIC Aztreonam (ATM) of 8 mg/L) According to Clinical Response by Infection Type at TOC: Aztreonam
Description: Population PK predicted (%fT>MIC ATM of 8 mg/L) for participants who received aztreonam-avibactam in studies C3601002 (NCT03329092) and C3601009 (NCT03580044). Clinical response categories included, clinical cure=improvement in baseline signs and symptoms such that after study treatment, no further antimicrobial treatment for the index infection (i.e., cIAI or HAP/VAP) was required. For cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. Failure was defined as participants who met any of the following criteria like death (after receiving at least 48 hours of study treatment) and participants who received treatment with further antibiotics for the index infection. Indeterminate was defined as death (after receiving less than 48 hours of study treatment) and for cIAI participants inadequate infection source control at time of initial surgical procedure.
Time Frame: At TOC (Day 28)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of time
Arm/Group | Aztreonam- Avibactam
Number analyzed (Participants) | 262
Percentage of time
  cIAI: Clinical cure: number analyzed (Participants) | 151
  cIAI: Clinical cure | 90.4 (41.9)
  cIAI: Failure: number analyzed (Participants) | 31
  cIAI: Failure | 73.81 (134.39)
  cIAI: Indeterminate: number analyzed (Participants) | 9
  cIAI: Indeterminate | 100 (0)
  HAP:Clinical cure: number analyzed (Participants) | 17
  HAP:Clinical cure | 97.87 (7.67)
  HAP: Failure: number analyzed (Participants) | 16
  HAP: Failure | 97.2 (8.4)
  HAP: Indeterminate: number analyzed (Participants) | 5
  HAP: Indeterminate | 100 (0)
  VAP: Clinical Cure: number analyzed (Participants) | 16
  VAP: Clinical Cure | 95.29 (8.94)
  VAP: Failure: number analyzed (Participants) | 16
  VAP: Failure | 96.38 (10.02)
  VAP: Indeterminate: number analyzed (Participants) | 1
  VAP: Indeterminate | 100 (NA) — SD was not estimated because of less number of participants in this events.

17. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over 24 Hours at Steady-state (AUC24,ss ) According to Clinical Response by Infection Type at TOC: Aztreonam
Description: Population PK predicted (AUC24,ss) for participants who received aztreonam-avibactam in studies C3601002 (NCT03329092) and C3601009 (NCT03580044). Clinical response categories included, clinical cure=improvement in baseline signs and symptoms such that after study treatment, no further antimicrobial treatment for the index infection (i.e., cIAI or HAP/VAP) was required. For cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. Failure was defined as participants who met any of the following criteria like death (after receiving at least 48 hours of study treatment) and participants who received treatment with further antibiotics for the index infection. Indeterminate was defined as death (after receiving less than 48 hours of study treatment) and for cIAI participants inadequate infection source control at time of initial surgical procedure.
Time Frame: 0 to 24 hours at TOC (Day 28)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligram*hours per liter (mg*h/L)
Arm/Group | Aztreonam- Avibactam
Number analyzed (Participants) | 262
Milligram*hours per liter (mg*h/L)
  cIAI: Clinical cure: number analyzed (Participants) | 151
  cIAI: Clinical cure | 816.18 (41.83)
  cIAI: Failure: number analyzed (Participants) | 31
  cIAI: Failure | 877.5 (85.91)
  cIAI: Indeterminate: number analyzed (Participants) | 9
  cIAI: Indeterminate | 1069.1 (15.82)
  HAP:Clinical cure: number analyzed (Participants) | 17
  HAP:Clinical cure | 1420.1 (54.62)
  HAP: Failure: number analyzed (Participants) | 16
  HAP: Failure | 1079.4 (34.1)
  HAP: Indeterminate: number analyzed (Participants) | 5
  HAP: Indeterminate | 1056.8 (35.68)
  VAP: Clinical cure: number analyzed (Participants) | 16
  VAP: Clinical cure | 858.39 (32.49)
  VAP: Failure: number analyzed (Participants) | 16
  VAP: Failure | 912.23 (38.1)
  VAP: Indeterminate: number analyzed (Participants) | 1
  VAP: Indeterminate | 1084.6 (NA) — SD was not estimated because of less number of participants in this events.

18. Secondary Outcome: Maximum Plasma Concentration for a Dosing Interval at Steady-state (Cmax,ss) According to Microbiological Response by Infection Type at TOC: Aztreonam
Description: Population PK predicted (Cmax,ss) for participants who received ATM-AVI in studies C3601002 (NCT03329092) and C3601009 (NCT03580044). Microbiological response included Favorable =baseline pathogens for participant had a favorable outcome. Eradication: Absence of causative pathogen from an appropriately obtained specimen at site of infection. Presumed eradication: repeat culture of specimens were not performed/clinically indicated in a participant who had a clinical response of cure. Unfavorable=persistence, persistence with increasing MIC, or presumed persistence. Persistence= Causative organism still present from appropriately obtained specimen at site of infection. Presumed persistence= Participant assessed as a clinical failure and repeat culture of specimens were not performed/clinically indicated. Indeterminate = death (after receiving < 48 hours of study treatment) and for cIAI participants inadequate infection source control at time of initial surgical procedure.
Time Frame: At TOC (Day 28)
Population: Analysis population included participants from PK and micro-ITT analysis set. All participants reported under 'Overall Number of Participants Analyzed' included participants evaluable for this outcome measure and contributed data to the table but may not have evaluable data for every row. Number Analyzed=participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligram per liter (mg/L)
Arm/Group | Aztreonam- Avibactam
Number analyzed (Participants) | 174
Milligram per liter (mg/L)
  cIAI: Favorable: number analyzed (Participants) | 108
  cIAI: Favorable | 53.26 (34.03)
  cIAI: Unfavorable: number analyzed (Participants) | 23
  cIAI: Unfavorable | 53.71 (67.14)
  cIAI: Indeterminate: number analyzed (Participants) | 4
  cIAI: Indeterminate | 62.97 (9.49)
  HAP:Favorable: number analyzed (Participants) | 8
  HAP:Favorable | 86.9 (71.56)
  HAP: Unfavorable: number analyzed (Participants) | 5
  HAP: Unfavorable | 55.48 (38.83)
  HAP: Indeterminate: number analyzed (Participants) | 3
  HAP: Indeterminate | 66.2 (33.87)
  VAP: Favorable: number analyzed (Participants) | 8
  VAP: Favorable | 50.71 (37.56)
  VAP: Unfavorable: number analyzed (Participants) | 14
  VAP: Unfavorable | 59.77 (31.52)
  VAP: Indeterminate: number analyzed (Participants) | 1
  VAP: Indeterminate | 85.34 (NA) — SD was not estimated because of less number of participants in this events.

19. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over 24 Hours at Steady-state (AUC24,ss) According to Microbiological Response by Infection Type at TOC: Aztreonam
Description: Population PK predicted (AUC24,ss) for participants who received ATM-AVI in studies C3601002 (NCT03329092) and C3601009 (NCT03580044). Microbiological response included Favorable =baseline pathogens for participant had a favorable outcome. Eradication: Absence of causative pathogen from an appropriately obtained specimen at site of infection. Presumed eradication: repeat culture of specimens were not performed/clinically indicated in a participant who had a clinical response of cure. Unfavorable=persistence, persistence with increasing MIC, or presumed persistence. Persistence= Causative organism still present from appropriately obtained specimen at site of infection. Presumed persistence= Participant assessed as a clinical failure and repeat culture of specimens were not performed/clinically indicated. Indeterminate = death (after receiving < 48 hours of study treatment) and for cIAI participants inadequate infection source control at time of initial surgical procedure.
Time Frame: 0 to 24 hours at TOC (Day 28)
Population: Analysis population included participants from PK and micro-ITT analysis set. All participants reported under 'Overall Number of Participants Analyzed' included participants evaluable for this outcome measure and contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' =participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligram*hours per liter
Arm/Group | Aztreonam- Avibactam
Number analyzed (Participants) | 174
Milligram*hours per liter
  cIAI: Favorable: number analyzed (Participants) | 108
  cIAI: Favorable | 830.23 (38.42)
  cIAI: Unfavorable: number analyzed (Participants) | 23
  cIAI: Unfavorable | 826.63 (95.22)
  cIAI: Indeterminate: number analyzed (Participants) | 4
  cIAI: Indeterminate | 1010.2 (9.17)
  HAP:Favorable: number analyzed (Participants) | 8
  HAP:Favorable | 1446.1 (82.6)
  HAP: Unfavorable: number analyzed (Participants) | 5
  HAP: Unfavorable | 909.59 (45.06)
  HAP: Indeterminate: number analyzed (Participants) | 3
  HAP: Indeterminate | 1237.9 (38.16)
  VAP: Favorable: number analyzed (Participants) | 8
  VAP: Favorable | 760.26 (40.54)
  VAP: Unfavorable: number analyzed (Participants) | 14
  VAP: Unfavorable | 974.21 (37.82)
  VAP: Indeterminate: number analyzed (Participants) | 1
  VAP: Indeterminate | 1084.6 (NA) — SD was not estimated because of less number of participants in this events.

20. Secondary Outcome: Percentage of Time That Free Plasma Concentrations Are Above the Minimum Inhibitory Concentration Over a Dosing Interval (%fT>MIC Aztreonam (ATM) of 8 mg/L) According to Microbiological Response by Infection Type at TOC: Aztreonam
Description: Population PK predicted (%fT>MIC ATM of 8 mg/L) for participants who received ATM-AVI in studies C3601002 (NCT03329092) and C3601009 (NCT03580044). Microbiological response included Favorable =baseline pathogens for participant had a favorable outcome. Eradication: Absence of causative pathogen from an appropriately obtained specimen at site of infection. Presumed eradication: repeat culture of specimens were not performed/clinically indicated in a participant who had a clinical response of cure. Unfavorable=persistence, persistence with increasing MIC, or presumed persistence. Persistence= Causative organism still present from appropriately obtained specimen at site of infection. Presumed persistence= Participant assessed as a clinical failure and repeat culture of specimens were not performed/clinically indicated. Indeterminate = death (after receiving < 48 hours of study treatment) and for cIAI participants inadequate infection source control at time of initial surgical procedure.
Time Frame: At TOC (Day 28)
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of time
Arm/Group | Aztreonam- Avibactam
Number analyzed (Participants) | 174
Percentage of time
  cIAI: Favorable: number analyzed (Participants) | 108
  cIAI: Favorable | 92.57 (17.66)
  cIAI: Unfavorable: number analyzed (Participants) | 23
  cIAI: Unfavorable | 68.02 (171.87)
  cIAI: Indeterminate: number analyzed (Participants) | 4
  cIAI: Indeterminate | 100 (0)
  HAP:Favorable: number analyzed (Participants) | 8
  HAP:Favorable | 95.53 (11.05)
  HAP: Unfavorable: number analyzed (Participants) | 5
  HAP: Unfavorable | 93.9 (14.14)
  HAP: Indeterminate: number analyzed (Participants) | 3
  HAP: Indeterminate | 100 (0)
  VAP: Favorable: number analyzed (Participants) | 8
  VAP: Favorable | 90.8 (12.3)
  VAP: Unfavorable: number analyzed (Participants) | 14
  VAP: Unfavorable | 97.42 (9.54)
  VAP: Indeterminate: number analyzed (Participants) | 1
  VAP: Indeterminate | 100 (NA) — SD was not estimated because of less number of participants in this events.

21. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over 24 Hours at Steady-state (AUC24,ss) According to Clinical Response by Infection Type at TOC: Avibactam
Description: as for outcome 17
Time Frame: 0 to 24 hours at TOC (Day 28)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligram*hour per liter
Arm/Group | Aztreonam- Avibactam
Number analyzed (Participants) | 262
Milligram*hour per liter
  cIAI: Clinical cure: number analyzed (Participants) | 151
  cIAI: Clinical cure | 164.92 (45.91)
  cIAI: Failure: number analyzed (Participants) | 31
  cIAI: Failure | 187.41 (96.93)
  cIAI: Indeterminate: number analyzed (Participants) | 9
  cIAI: Indeterminate | 213.92 (20.81)
  HAP:Clinical cure: number analyzed (Participants) | 17
  HAP:Clinical cure | 291.47 (61.75)
  HAP: Failure: number analyzed (Participants) | 16
  HAP: Failure | 214.99 (36.09)
  HAP: Indeterminate: number analyzed (Participants) | 5
  HAP: Indeterminate | 257.37 (71.75)
  VAP: Clinical cure: number analyzed (Participants) | 16
  VAP: Clinical cure | 176.95 (31.43)
  VAP: Failure: number analyzed (Participants) | 16
  VAP: Failure | 178.68 (38.99)
  VAP: Indeterminate: number analyzed (Participants) | 1
  VAP: Indeterminate | 218.09 (NA) — SD was not estimated because of less number of participants in this events.

22. Secondary Outcome: Maximum Plasma Concentration for a Dosing Interval at Steady-state (Cmax,ss ) According to Clinical Response by Infection Type at TOC: Avibactam
Description: Population PK predicted (Cmax,ss) for participants who received aztreonam-avibactam in studies C3601002 (NCT03329092) and C3601009 (NCT03580044). Clinical response categories included, clinical cure=improvement in baseline signs and symptoms such that after study treatment, no further antimicrobial treatment for the index infection (i.e., cIAI or HAP/VAP) was required. For cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. Failure was defined as participants who met any of the following criteria like death (after receiving at least 48 hours of study treatment) and participants who received treatment with further antibiotics for the index infection. Indeterminate was defined as death (after receiving less than 48 hours of study treatment) and for cIAI participants inadequate infection source control at time of initial surgical procedure.
Time Frame: At TOC (Day 28)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligram per liter (mg/L)
Arm/Group | Aztreonam- Avibactam
Number analyzed (Participants) | 262
Milligram per liter (mg/L)
  cIAI: Clinical cure: number analyzed (Participants) | 151
  cIAI: Clinical cure | 11.01 (42.14)
  cIAI: Failure: number analyzed (Participants) | 31
  cIAI: Failure | 12.48 (72.59)
  cIAI: Indeterminate: number analyzed (Participants) | 9
  cIAI: Indeterminate | 14.04 (16.52)
  HAP:Clinical cure: number analyzed (Participants) | 17
  HAP:Clinical cure | 18.41 (55.07)
  HAP: Failure: number analyzed (Participants) | 16
  HAP: Failure | 13.46 (33.52)
  HAP: Indeterminate: number analyzed (Participants) | 5
  HAP: Indeterminate | 15.24 (49.1)
  VAP: Clinical Cure: number analyzed (Participants) | 16
  VAP: Clinical Cure | 11.64 (31.01)
  VAP: Failure: number analyzed (Participants) | 16
  VAP: Failure | 11.44 (32.65)
  VAP: Indeterminate: number analyzed (Participants) | 1
  VAP: Indeterminate | 18.93 (NA) — SD was not estimated because of less number of participants in this events.

23. Secondary Outcome: Percent of Time That Free Plasma Concentrations Are Above the Threshold Concentration Over a Dosing Interval (%fT>CT of 2.5mg/L) According to Clinical Response by Infection Type at TOC: Avibactam
Description: Population PK predicted (%fT>CT of 2.5mg/L) for participants who received aztreonam-avibactam in studies C3601002 (NCT03329092) and C3601009 (NCT03580044). Clinical response categories included, clinical cure=improvement in baseline signs and symptoms such that after study treatment, no further antimicrobial treatment for the index infection (i.e., cIAI or HAP/VAP) was required. For cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. Failure was defined as participants who met any of the following criteria like death (after receiving at least 48 hours of study treatment) and participants who received treatment with further antibiotics for the index infection. Indeterminate was defined as death (after receiving less than 48 hours of study treatment) and for cIAI participants inadequate infection source control at time of initial surgical procedure.
Time Frame: At TOC (Day 28)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of time
Arm/Group | Aztreonam- Avibactam
Number analyzed (Participants) | 262
Percentage of time
  cIAI: Clinical cure: number analyzed (Participants) | 151
  cIAI: Clinical cure | 85.53 (43.26)
  cIAI: Failure: number analyzed (Participants) | 31
  cIAI: Failure | 71.92 (133.68)
  cIAI: Indeterminate: number analyzed (Participants) | 9
  cIAI: Indeterminate | 98.52 (2.81)
  HAP:Clinical cure: number analyzed (Participants) | 17
  HAP:Clinical cure | 95.99 (11.57)
  HAP: Failure: number analyzed (Participants) | 16
  HAP: Failure | 95.28 (12.12)
  HAP: Indeterminate: number analyzed (Participants) | 5
  HAP: Indeterminate | 92.75 (11.19)
  VAP: Clinical Cure: number analyzed (Participants) | 16
  VAP: Clinical Cure | 92 (13.01)
  VAP: Failure: number analyzed (Participants) | 16
  VAP: Failure | 94.08 (12.93)
  VAP: Indeterminate: number analyzed (Participants) | 1
  VAP: Indeterminate | 100 (NA) — SD was not estimated because of less number of participants in this events.

24. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over 24 Hours at Steady-state (AUC24,ss) According to Microbiological Response by Infection Type at TOC: Avibactam
Description: Population PK predicted (AUC24,ss) for participants who received ATM-AVI in studies C3601002 (NCT03329092) and C3601009 (NCT03580044). Microbiological response included Favorable =baseline pathogens for participant had a favorable outcome. Eradication: Absence of causative pathogen from an appropriately obtained specimen at site of infection. Presumed eradication: repeat culture of specimens were not performed/clinically indicated in a participant who had a clinical response of cure. Unfavorable=persistence, persistence with increasing MIC, or presumed persistence. Persistence= Causative organism still present from appropriately obtained specimen at site of infection. Presumed persistence= Participant assessed as a clinical failure and repeat culture of specimens were not performed/clinically indicated. Indeterminate = death (after receiving<48 hours of study treatment) and for cIAI participants inadequate infection source control at time of initial surgical procedure.
Time Frame: 0 to 24 hours At TOC (Day 28)
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligram*hours per liter
Arm/Group | Aztreonam- Avibactam
Number analyzed (Participants) | 174
Milligram*hours per liter
  cIAI: Favorable: number analyzed (Participants) | 108
  cIAI: Favorable | 166.4 (40.88)
  cIAI: Unfavorable: number analyzed (Participants) | 23
  cIAI: Unfavorable | 177.65 (106.25)
  cIAI: Indeterminate: number analyzed (Participants) | 4
  cIAI: Indeterminate | 197.01 (7.31)
  HAP:Favorable: number analyzed (Participants) | 8
  HAP:Favorable | 293.49 (95.13)
  HAP: Unfavorable: number analyzed (Participants) | 5
  HAP: Unfavorable | 196.38 (61.95)
  HAP: Indeterminate: number analyzed (Participants) | 3
  HAP: Indeterminate | 359.31 (71.12)
  VAP: Favorable: number analyzed (Participants) | 8
  VAP: Favorable | 157.79 (43.71)
  VAP: Unfavorable: number analyzed (Participants) | 14
  VAP: Unfavorable | 192.85 (38.42)
  VAP: Indeterminate: number analyzed (Participants) | 1
  VAP: Indeterminate | 218.09 (NA) — SD was not estimated because of less number of participants in this events.

25. Secondary Outcome: Maximum Plasma Concentration for a Dosing Interval at Steady-state (Cmax,ss (mg/L)) According to Microbiological Response by Infection Type at TOC: Avibactam
Description: Population PK predicted (Cmax,ss (mg/L)) for participants who received ATM-AVI in studies C3601002 (NCT03329092) and C3601009 (NCT03580044). Microbiological response included Favorable =baseline pathogens for participant had a favorable outcome. Eradication: Absence of causative pathogen from an appropriately obtained specimen at site of infection. Presumed eradication: repeat culture of specimens were not performed/clinically indicated in a participant who had a clinical response of cure. Unfavorable=persistence, persistence with increasing MIC, or presumed persistence. Persistence= Causative organism still present from appropriately obtained specimen at site of infection. Presumed persistence= Participant assessed as a clinical failure and repeat culture of specimens were not performed/clinically indicated. Indeterminate = death (after receiving<48 hours of study treatment) and for cIAI participants inadequate infection source control at time of initial surgical procedure.
Time Frame: At TOC (Day 28)
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligram per liter (mg/L)
Arm/Group | Aztreonam- Avibactam
Number analyzed (Participants) | 174
Milligram per liter (mg/L)
  cIAI: Favorable: number analyzed (Participants) | 108
  cIAI: Favorable | 11.1 (37.2)
  cIAI: Unfavorable: number analyzed (Participants) | 23
  cIAI: Unfavorable | 11.83 (76.48)
  cIAI: Indeterminate: number analyzed (Participants) | 4
  cIAI: Indeterminate | 13.03 (8.01)
  HAP:Favorable: number analyzed (Participants) | 8
  HAP:Favorable | 18.55 (84.68)
  HAP: Unfavorable: number analyzed (Participants) | 5
  HAP: Unfavorable | 12.31 (51.34)
  HAP: Indeterminate: number analyzed (Participants) | 3
  HAP: Indeterminate | 18.72 (55.03)
  VAP: Favorable: number analyzed (Participants) | 8
  VAP: Favorable | 10.75 (42.72)
  VAP: Unfavorable: number analyzed (Participants) | 14
  VAP: Unfavorable | 12.28 (32.85)
  VAP: Indeterminate: number analyzed (Participants) | 1
  VAP: Indeterminate | 18.93 (NA) — SD was not estimated because of less number of participants in this events.

26. Secondary Outcome: Percent of Time That Free Plasma Concentrations Are Above the Threshold Concentration Over a Dosing Interval; (%fT>CT of 2.5 mg/L) According to Microbiological Response by Infection Type at TOC: Avibactam
Description: Population PK predicted (%fT>CT of 2.5 mg/L) for participants who received ATM-AVI in studies C3601002 (NCT03329092) and C3601009 (NCT03580044). Microbiological response included Favorable =baseline pathogens for participant had a favorable outcome. Eradication: Absence of causative pathogen from an appropriately obtained specimen at site of infection. Presumed eradication: repeat culture of specimens were not performed/clinically indicated in a participant who had a clinical response of cure. Unfavorable=persistence, persistence with increasing MIC, or presumed persistence. Persistence= Causative organism still present from appropriately obtained specimen at site of infection. Presumed persistence= Participant assessed as a clinical failure and repeat culture of specimens were not performed/clinically indicated. Indeterminate = death (after receiving < 48 hours of study treatment) and for cIAI participants inadequate infection source control at time of initial surgical procedure.
Time Frame: At TOC (Day 28)
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of time
Groups:
- Avibactam: Participants who received AVI in studies C3601002 (NCT03329092) and C3601009 (NCT03580044) were included in the analysis.
Arm/Group | Avibactam
Number analyzed (Participants) | 174
Percentage of time
  cIAI: Favorable: number analyzed (Participants) | 108
  cIAI: Favorable | 87.93 (21.78)
  cIAI: Unfavorable: number analyzed (Participants) | 23
  cIAI: Unfavorable | 66.43 (170.59)
  cIAI: Indeterminate: number analyzed (Participants) | 4
  cIAI: Indeterminate | 99.24 (1.52)
  HAP:Favorable: number analyzed (Participants) | 8
  HAP:Favorable | 92.26 (16.44)
  HAP: Unfavorable: number analyzed (Participants) | 5
  HAP: Unfavorable | 90.03 (18.83)
  HAP: Indeterminate: number analyzed (Participants) | 3
  HAP: Indeterminate | 100 (0)
  VAP: Favorable: number analyzed (Participants) | 8
  VAP: Favorable | 87.47 (16.8)
  VAP: Unfavorable: number analyzed (Participants) | 14
  VAP: Unfavorable | 95.52 (11.79)
  VAP: Indeterminate: number analyzed (Participants) | 1
  VAP: Indeterminate | 100 (NA) — SD was not estimated because of less number of participants in this events.

27. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs
Description: An adverse event (AE) was any untoward medical occurrence in a study participant administered medicinal product,; the event need not necessarily have a causal relationship with product treatment or usage. A serious adverse event (SAE) was any untoward medical occurrence at any dose that: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital abnormal/birth defect or considered an important medical event.
Time Frame: From start of study treatment until end of late follow-up (Up to Day 45)
Population: Safety analysis set included all participants who received any amount of study treatment. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 275 | 137
Participants
  AEs | 177 | 87
  SAEs | 53 | 25

28. Secondary Outcome: Number of Participants With Potentially Clinically Significant Hematology Abnormalities
Description: Criteria for potential clinically significant hematology results were as follows: hemoglobin, hematocrit and erythrocyte <0.7*lower limit of normal [LLN] and >30% decrease from Baseline (DFB); >1.3*upper limit of normal (ULN) and >30% increase from Baseline (IFB). Platelet count <0.65*LLN and > 50% decrease from baseline; > 1.5 * ULN and > 100% increase from baseline. leukocyte: < 0.65* LLN and > 60% decrease from baseline; > 1.5* ULN and 100% increase from baseline. Neutrophils/leukocytes < 0.65 * LLN and >75% decrease from baseline; > 1.6*ULN and > 100% increase from baseline. Lymphocytes/leukocytes < 0.25* LLN and > 75% decrease from baseline;> 1.5* ULN and > 100% increase from baseline, Eosinophils/leukocytes, Monocytes/leukocytes, Basophils/leukocytes > 4.0* ULN and > 300% increase from baseline.
Time Frame: From start of study treatment until TOC visit (Up to Day 28)
Population: Safety analysis set included all participants who received any amount of study treatment. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants available for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 275 | 137
Participants
  Hematocrit < 0.7*LLN and > 30% Decrease from Baseline: number analyzed (Participants) | 258 | 127
  Hematocrit < 0.7*LLN and > 30% Decrease from Baseline | 6 | 3
  Hematocrit > 1.3* ULN and > 30% Increase from Baseline: number analyzed (Participants) | 258 | 127
  Hematocrit > 1.3* ULN and > 30% Increase from Baseline | 0 | 0
  Hemoglobin< 0.7* LLN and > 30% Decrease from Baseline: number analyzed (Participants) | 259 | 133
  Hemoglobin< 0.7* LLN and > 30% Decrease from Baseline | 8 | 3
  Hemoglobin > 1.3* ULN and > 30% Increase from Baseline: number analyzed (Participants) | 259 | 133
  Hemoglobin > 1.3* ULN and > 30% Increase from Baseline | 0 | 0
  Erythrocytes < 0.7* LLN and > 30% Decrease from Baseline: number analyzed (Participants) | 259 | 133
  Erythrocytes < 0.7* LLN and > 30% Decrease from Baseline | 7 | 3
  Erythrocytes > 1.3* ULN and > 30% Increase from Baseline: number analyzed (Participants) | 259 | 133
  Erythrocytes > 1.3* ULN and > 30% Increase from Baseline | 0 | 0
  Leukocytes < 0.65* LLN and > 60% Decrease from Baseline: number analyzed (Participants) | 260 | 133
  Leukocytes < 0.65* LLN and > 60% Decrease from Baseline | 0 | 0
  Leukocytes > 1.5* ULN and > 100% Increase from Baseline: number analyzed (Participants) | 260 | 133
  Leukocytes > 1.5* ULN and > 100% Increase from Baseline | 12 | 5
  Neutrophils/Leukocytes < 0.65* LLN and > 75% Decrease from Baseline: number analyzed (Participants) | 259 | 131
  Neutrophils/Leukocytes < 0.65* LLN and > 75% Decrease from Baseline | 0 | 0
  Neutrophils/Leukocytes > 1.6* ULN and > 100% Increase from Baseline: number analyzed (Participants) | 259 | 131
  Neutrophils/Leukocytes > 1.6* ULN and > 100% Increase from Baseline | 0 | 0
  Monocytes/Leukocytes > 4.0* ULN and > 300% Increase from Baseline: number analyzed (Participants) | 258 | 131
  Monocytes/Leukocytes > 4.0* ULN and > 300% Increase from Baseline | 0 | 0
  Lymphocytes/Leukocytes < 0.25* LLN and > 75% Decrease from Baseline: number analyzed (Participants) | 258 | 132
  Lymphocytes/Leukocytes < 0.25* LLN and > 75% Decrease from Baseline | 1 | 1
  Lymphocytes/Leukocytes > 1.5* ULN and > 100% Increase from Baseline: number analyzed (Participants) | 258 | 132
  Lymphocytes/Leukocytes > 1.5* ULN and > 100% Increase from Baseline | 0 | 0
  Eosinophils/Leukocytes > 4.0* ULN and > 300% Increase from Baseline: number analyzed (Participants) | 258 | 131
  Eosinophils/Leukocytes > 4.0* ULN and > 300% Increase from Baseline | 0 | 0
  Basophils/Leukocytes > 4.0* ULN and > 300% Increase from Baseline: number analyzed (Participants) | 258 | 131
  Basophils/Leukocytes > 4.0* ULN and > 300% Increase from Baseline | 0 | 0
  Platelets < 0.65* LLN and > 50% Decrease from Baseline: number analyzed (Participants) | 259 | 131
  Platelets < 0.65* LLN and > 50% Decrease from Baseline | 3 | 2
  Platelets > 1.5* ULN and > 100% Increase from Baseline: number analyzed (Participants) | 259 | 131
  Platelets > 1.5* ULN and > 100% Increase from Baseline | 12 | 7

29. Secondary Outcome: Number of Participants With Potentially Clinically Significant Clinical Chemistry Abnormalities
Description: Albumin < 0.5* LLN and> 50% decrease from baseline (DFB);> 1.5 * ULN and> 50% increase from baseline (IFB). Alkaline phosphatase < 0.5 * LLN and> 80% DFB;> 3.0 * ULN and> 100%. Alanine and Aspartate aminotransferase > 3.0 * ULN and> 100% IFB. Bicarbonate < 0.7 * LLN and > 40% DFB;> 1.3 * ULN and> 40% IFB. Blood urea nitrogen < 0.2 * LLN and > 100% DFB; > 3.0 * ULN and > 200% IFB. Calcium < 0.7 * LLN and > 30% DFB;> 1.3 * ULN and> 30% IFB. Chloride < 0.8 * LLN >and 20% DFB; > 1.2 * ULN and > 20% IFB. Creatinine > 2.0 * ULN and> 100% IFB; Glucose < 0.6 * LLN and> 40% DFB; > 3.0 * ULN and> 200% IFB. Potassium < 0.8 * LLN and > 20% DFB; > 1.2 * ULN and> 20% IFB. Sodium < 0.85 * LLN and> 10% DFB;> 1.1 * ULN and >10% IFB. Bilirubin > 1.5 * ULN and > 100% IFB.; Direct bilirubin > 2.0 * ULN and > 150% IFB.
Time Frame: From start of study treatment until At TOC visit (Up to Day 28)
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 275 | 137
Participants
  Aspartate Aminotransferase >3.0* ULN and > 100% Increase from Baseline: number analyzed (Participants) | 262 | 133
  Aspartate Aminotransferase >3.0* ULN and > 100% Increase from Baseline | 25 | 14
  Alanine Aminotransferase > 3.0* ULN and > 100% Increase from Baseline: number analyzed (Participants) | 264 | 132
  Alanine Aminotransferase > 3.0* ULN and > 100% Increase from Baseline | 24 | 10
  Alkaline Phosphatase < 0.5* LLN and > 80% Decrease from Baseline: number analyzed (Participants) | 264 | 133
  Alkaline Phosphatase < 0.5* LLN and > 80% Decrease from Baseline | 0 | 0
  Alkaline Phosphatase > 3.0* ULN and > 100% Increase from Baseline: number analyzed (Participants) | 264 | 133
  Alkaline Phosphatase > 3.0* ULN and > 100% Increase from Baseline | 5 | 4
  Bilirubin > 1.5* ULN and > 100% Increase from Baseline: number analyzed (Participants) | 263 | 132
  Bilirubin > 1.5* ULN and > 100% Increase from Baseline | 2 | 3
  Direct Bilirubin > 2.0* ULN and > 150% Increase from Baseline: number analyzed (Participants) | 258 | 130
  Direct Bilirubin > 2.0* ULN and > 150% Increase from Baseline | 2 | 0
  Creatinine > 2.0* ULN and > 100% Increase from Baseline: number analyzed (Participants) | 270 | 136
  Creatinine > 2.0* ULN and > 100% Increase from Baseline | 0 | 3
  Sodium < 0.85* LLN and > 10% Decrease from Baseline: number analyzed (Participants) | 263 | 133
  Sodium < 0.85* LLN and > 10% Decrease from Baseline | 0 | 0
  Sodium> 1.1* ULN and > 10% Increase from Baseline: number analyzed (Participants) | 263 | 133
  Sodium> 1.1* ULN and > 10% Increase from Baseline | 0 | 0
  Potassium < 0.8* LLN and > 20% Decrease from Baseline: number analyzed (Participants) | 262 | 132
  Potassium < 0.8* LLN and > 20% Decrease from Baseline | 6 | 1
  Potassium > 1.2* ULN and > 20% Increase from Baseline: number analyzed (Participants) | 262 | 132
  Potassium > 1.2* ULN and > 20% Increase from Baseline | 5 | 4
  Chloride< 0.8* LLN and > 20% Decrease from Baseline: number analyzed (Participants) | 263 | 133
  Chloride< 0.8* LLN and > 20% Decrease from Baseline | 0 | 0
  Chloride > 1.2* ULN and > 20% Increase from Baseline: number analyzed (Participants) | 263 | 133
  Chloride > 1.2* ULN and > 20% Increase from Baseline | 1 | 0
  Bicarbonate < 0.7* LLN and > 40% Decrease from Baseline: number analyzed (Participants) | 257 | 129
  Bicarbonate < 0.7* LLN and > 40% Decrease from Baseline | 0 | 0
  Bicarbonate > 1.3* ULN and > 40% Increase from Baseline: number analyzed (Participants) | 257 | 129
  Bicarbonate > 1.3* ULN and > 40% Increase from Baseline | 3 | 1
  Calcium < 0.7* LLN and > 30% Decrease from Baseline: number analyzed (Participants) | 262 | 130
  Calcium < 0.7* LLN and > 30% Decrease from Baseline | 2 | 1
  Calcium > 1.3* ULN and > 30% Increase from Baseline: number analyzed (Participants) | 262 | 130
  Calcium > 1.3* ULN and > 30% Increase from Baseline | 0 | 0
  Albumin < 0.5* LLN and > 50% Decrease from Baseline: number analyzed (Participants) | 261 | 132
  Albumin < 0.5* LLN and > 50% Decrease from Baseline | 0 | 0
  Albumin > 1.5* ULN and > 50% Increase from Baseline: number analyzed (Participants) | 261 | 132
  Albumin > 1.5* ULN and > 50% Increase from Baseline | 0 | 0
  Glucose < 0.6* LLN and > 40% Decrease from Baseline: number analyzed (Participants) | 261 | 132
  Glucose < 0.6* LLN and > 40% Decrease from Baseline | 0 | 1
  Glucose > 3.0* ULN and > 200% Increase from Baseline: number analyzed (Participants) | 261 | 132
  Glucose > 3.0* ULN and > 200% Increase from Baseline | 2 | 0
  Urea Nitrogen < 0.2* LLN and > 100% Decrease from Baseline: number analyzed (Participants) | 259 | 130
  Urea Nitrogen < 0.2* LLN and > 100% Decrease from Baseline | 0 | 0
  Urea Nitrogen > 3.0* ULN and > 200% Increase from Baseline: number analyzed (Participants) | 259 | 130
  Urea Nitrogen > 3.0* ULN and > 200% Increase from Baseline | 0 | 0

30. Secondary Outcome: Number of Participants With Abnormalities in Vital Signs
Description: Vitals signs, included blood pressure and, heart rate. Blood pressure (BP) and heart rate were measured using a semiautomatic BP recording device with the participant in a supine position after at least 10 minutes of rest. Criteria for abnormalities included: Systolic BP (millimeters of mercury [mmHg]): value more than (>) 150 and increase from baseline more than equal (>= 30) or value less than (<) 90 and decrease from baseline >= 30; DBP: value > 100 and increase from baseline >=20 or Value < 50 and decrease from baseline >= 20; Heart Rate (beats per minute [BPM]): value < 40 or > 120.
Time Frame: From start of study treatment until TOC visit (Up to Day 28)
Population: Safety analysis set included all participants who received any amount of study treatment. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 271 | 136
Participants
  Systolic BP (mmHg) Value more than (>) 150 and increase from baseline more than equal (≥ to 30) | 35 | 16
  Systolic BP (mmHg) Value less than (<) 90 and decrease from baseline more than equal (≥) 30 | 8 | 3
  Diastolic BP (mmHg) Value > 100 and increase from baseline ≥ 20 | 8 | 0
  Diastolic BP (mmHg) Value < 50 and decrease from baseline ≥ 20 | 10 | 5
  Heart Rate (BPM) Value < 40 or > 120: number analyzed (Participants) | 270 | 136
  Heart Rate (BPM) Value < 40 or > 120 | 265 | 135

31. Secondary Outcome: Number of Participants With Abnormal Physical Examination Finding
Description: A complete physical examination was performed and included an assessment of the following: general appearance including site of infection, skin, head and throat (head, eyes, ears, nose, and throat), lymph nodes, lungs, cardiovascular (CV), abdomen, musculoskeletal, and neurological systems.
Time Frame: Screening, End of treatment (up to 24 hours post infusion on Day 14) and Test of Cure (Day 28)
Population: The safety analysis set included all participants who received any amount of study treatment. Here, 'Number Analyzed' signifies number of participants available for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 275 | 137
Participants
  Abdomen: Screening | 184 | 103
  Abdomen: End of Treatment: number analyzed (Participants) | 263 | 130
  Abdomen: End of Treatment | 56 | 30
  Abdomen: Test of Cure: number analyzed (Participants) | 230 | 112
  Abdomen: Test of Cure | 31 | 12
  Cardiovascular: Screening | 50 | 22
  Cardiovascular: End of Treatment: number analyzed (Participants) | 264 | 129
  Cardiovascular: End of Treatment | 27 | 14
  Cardiovascular: Test of Cure: number analyzed (Participants) | 230 | 113
  Cardiovascular: Test of Cure | 20 | 10
  Ears: Screening: number analyzed (Participants) | 270 | 137
  Ears: Screening | 1 | 1
  Ears: End of Treatment: number analyzed (Participants) | 261 | 128
  Ears: End of Treatment | 0 | 1
  Ears:Test of Cure: number analyzed (Participants) | 228 | 112
  Ears:Test of Cure | 0 | 1
  Eyes: Screening: number analyzed (Participants) | 272 | 137
  Eyes: Screening | 13 | 4
  Eyes End of Treatment: number analyzed (Participants) | 262 | 128
  Eyes End of Treatment | 7 | 1
  Eyes: Test of Cure: number analyzed (Participants) | 228 | 112
  Eyes: Test of Cure | 6 | 1
  General appearance: Screening: number analyzed (Participants) | 273 | 137
  General appearance: Screening | 77 | 35
  General appearance: End of Treatment: number analyzed (Participants) | 263 | 129
  General appearance: End of Treatment | 34 | 15
  General appearance: Test of Cure: number analyzed (Participants) | 228 | 113
  General appearance: Test of Cure | 16 | 8
  Head: Screening: number analyzed (Participants) | 271 | 136
  Head: Screening | 12 | 4
  Head: End of Treatment: number analyzed (Participants) | 263 | 127
  Head: End of Treatment | 10 | 5
  Head: Test of Cure: number analyzed (Participants) | 229 | 111
  Head: Test of Cure | 6 | 2
  Lungs: Screening | 70 | 37
  Lungs: End of Treatment: number analyzed (Participants) | 264 | 129
  Lungs: End of Treatment | 45 | 15
  Lungs: Test of Cure: number analyzed (Participants) | 231 | 113
  Lungs: Test of Cure | 22 | 8
  Lymph nodes: Screening: number analyzed (Participants) | 271 | 136
  Lymph nodes: Screening | 1 | 0
  Lymph nodes: End of Treatment: number analyzed (Participants) | 258 | 128
  Lymph nodes: End of Treatment | 1 | 0
  Lymph nodes: Test of Cure: number analyzed (Participants) | 228 | 112
  Lymph nodes: Test of Cure | 0 | 0
  Musculoskeletal: Screening | 21 | 10
  Musculoskeletal: End of Treatment: number analyzed (Participants) | 262 | 129
  Musculoskeletal: End of Treatment | 17 | 9
  Musculoskeletal: Test of Cure: number analyzed (Participants) | 228 | 112
  Musculoskeletal: Test of Cure | 9 | 3
  Neurological: Screening: number analyzed (Participants) | 273 | 136
  Neurological: Screening | 37 | 13
  Neurological: End of Treatment: number analyzed (Participants) | 262 | 130
  Neurological: End of Treatment | 34 | 9
  Neurological: Test of Cure: number analyzed (Participants) | 229 | 112
  Neurological: Test of Cure | 17 | 6
  Nose: Screening: number analyzed (Participants) | 271 | 137
  Nose: Screening | 4 | 3
  Nose: End of Treatment: number analyzed (Participants) | 262 | 128
  Nose: End of Treatment | 2 | 0
  Nose: Test of Cure: number analyzed (Participants) | 228 | 112
  Nose: Test of Cure | 1 | 0
  Skin: Screening: number analyzed (Participants) | 274 | 137
  Skin: Screening | 47 | 25
  Skin: End of Treatment: number analyzed (Participants) | 262 | 129
  Skin: End of Treatment | 33 | 22
  Skin: Test of Cure: number analyzed (Participants) | 229 | 113
  Skin: Test of Cure | 21 | 12
  Throat: Screening: number analyzed (Participants) | 266 | 136
  Throat: Screening | 9 | 0
  Throat: End of Treatment: number analyzed (Participants) | 258 | 128
  Throat: End of Treatment | 10 | 1
  Throat: Test of Cure: number analyzed (Participants) | 227 | 111
  Throat: Test of Cure | 4 | 1

32. Secondary Outcome: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Findings
Description: Standard 12-lead ECGs were recorded with the participants in the supine position after the participant had rested in this position for 10 minutes. Clinically significant findings were based on investigators assessment.
Time Frame: Baseline (latest non-missing value before start of treatment) and Day 3
Population: The safety analysis set included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 275 | 137
Participants
  Baseline | 16 | 5
  Day 3 | 11 | 6

33. Other Pre Specified Outcome: Percentage of Participants With Clinical Cure at End of Treatment (EOT) Visit: ITT Analysis Set
Description: as for outcome 3
Time Frame: At EOT visit (Within 24 hours after last infusion on Day 14)
Population: The ITT analysis set included all randomized participants regardless of the treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 282 | 140
Percentage of participants | 75.9 [70.6 to 80.6] | 73.6 [65.8 to 80.3]
Statistical Analysis 1: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; Test type: Other; Difference in clinical cure rate = 2.3, 95% CI 2-sided [-6.2 to 11.5] — CI for the difference was calculated using the unstratified Miettinen and Nurminen method

34. Other Pre Specified Outcome: Percentage of Participants With Clinical Cure at EOT Visit: Micro-ITT Analysis Set
Description: Clinical cure was defined as improvement in baseline signs and symptoms such that after study treatment, no further antimicrobial treatment for the index infection (i.e., cIAI or HAP/VAP) was required. For cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. Clinical cure was determined by the Independent Clinical Adjudication Committee. 95% CI was based on Jeffrey's method.
Time Frame: At EOT visit (Within 24 hours after last infusion on Day 14)
Population: Micro-ITT analysis set was a subset of the ITT analysis set and included all participants who had at least one Gram-negative baseline pathogen from an adequate specimen obtained prior to the start of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Meropenem± Colistimethate: Participants hospitalized with cIAI or NP (including HAP and VAP) were randomized to receive 1000 mg meropenem every 8 hours by IV infusion. A higher dose of 2000 mg was given by IV infusion over 180 minutes carbapenem resistant pathogen was strongly suspected. Participants were administered colistimethate sodium at investigator's discretion.
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 177 | 94
Percentage of participants | 79.7 [73.3 to 85.1] | 80.9 [72.0 to 87.8]
Statistical Analysis 1: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; Test type: Other; Difference in clinical cure = -1.2, 95% CI 2-sided [-10.7 to 9.4] — CI for the difference was calculated using the unstratified Miettinen and Nurminen method

35. Other Pre Specified Outcome: Percentage of Participants With Clinical Cure at EOT Visit: CE Analysis Set
Description: Clinical cure = improvement in baseline signs and symptoms such that after study treatment, no further antimicrobial treatment for the index infection (i.e., cIAI or HAP/VAP) was required. Additionally, for cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. Clinical cure was determined by the Independent Clinical Adjudication Committee. 95% CI was based on Jeffrey's method. CE analysis set: all participants in ITT analysis set; met criteria for cIAI, or HAP/VAP; received at least 48 hours of study treatment or <48 hours of treatment before discontinuing study drug due to AE; no concomitant antibiotics for any baseline pathogens between first dose and TOC (except protocol-allowed antibiotics); no prior antibiotics other than allowed per protocol; no important protocol deviations; no clinical outcome of indeterminate at TOC; no monomicrobial infections due to non-eligible pathogens and did not have only Gram-positive pathogens.
Time Frame: At EOT visit (Within 24 hours after last infusion on Day 14)
Population: Analysis was performed on CE analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 213 | 105
Percentage of participants | 82.2 [76.6 to 86.8] | 81.9 [73.7 to 88.4]
Statistical Analysis 1: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; Test type: Other; Difference in clinical cure = 0.3, 95% CI 2-sided [-8.3 to 9.9] — CI for the difference was calculated using the unstratified Miettinen and Nurminen method

36. Other Pre Specified Outcome: Percentage of Participants With Clinical Cure at EOT Visit: ME Analysis Set
Description: as for outcome 3
Time Frame: At EOT visit (Within 24 hours after last infusion on Day 14)
Population: The ME analysis set included all participants commonly included in both micro-ITT and CE analysis sets and included participants who have at least 1 etiologic pathogen from an adequate baseline culture regardless of susceptibility to study agents.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 149 | 79
Percentage of participants | 84.6 [78.1 to 89.7] | 83.5 [74.2 to 90.4]
Statistical Analysis 1: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; Test type: Other; Difference in clinical cure rate = 1.0, 95% CI 2-sided [-8.5 to 12.0] — CI for the difference was calculated using the unstratified Miettinen and Nurminen method

37. Other Pre Specified Outcome: Percentage of Participants With Clinical Cure by Type of Infection at EOT Visit: ITT Analysis Set
Description: as for outcome 3
Time Frame: At EOT visit (Within 24 hours after last infusion on Day 14)
Population: The ITT analysis set included all randomized participants regardless of the treatment received. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 282 | 140
Percentage of participants
  cIAI: number analyzed (Participants) | 208 | 104
  cIAI | 81.7 [76.1 to 86.5] | 79.8 [71.3 to 86.6]
  HAP/VAP: number analyzed (Participants) | 74 | 36
  HAP/VAP | 59.5 [48.1 to 70.1] | 55.6 [39.4 to 70.8]
Statistical Analysis 1: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; cIAI; Test type: Other; Difference in clinical cure rate = 1.9, 95% CI 2-sided [-6.9 to 11.9] — CI for the difference was calculated using the unstratified Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; HAP/VAP; Test type: Other; Difference in clinical cure rate = 3.9, 95% CI 2-sided [-15.2 to 23.4] — CI for the difference was calculated using the unstratified Miettinen and Nurminen method

38. Other Pre Specified Outcome: Percentage of Participants With Clinical Cure by Type of Infection at EOT Visit: CE Analysis Set
Description: as for outcome 35
Time Frame: At EOT visit (Within 24 hours after last infusion on Day 24)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 213 | 105
Percentage of participants
  cIAI: number analyzed (Participants) | 168 | 83
  cIAI | 88.7 [83.2 to 92.8] | 85.5 [76.8 to 91.8]
  HAP/VAP: number analyzed (Participants) | 45 | 22
  HAP/VAP | 57.8 [43.2 to 71.4] | 68.2 [47.4 to 84.5]
Statistical Analysis 1: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; cIAI; Test type: Other; Difference in clinical cure rate = 3.1, 95% CI 2-sided [-5.2 to 13.2] — CI for the difference was calculated using the unstratified Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Aztreonam-avibactam ± Metronidazole vs Meropenem± Colistimethate; HAP/VAP; Test type: Other; Difference in clinical cure rate = -10.4, 95% CI 2-sided [-32.6 to 14.9] — CI for the difference was calculated using the unstratified Miettinen and Nurminen method

39. Other Pre Specified Outcome: Percentage of Participants With Clinical Cure by Pathogen Resistance Type at EOT Visit: Micro-ITT Analysis Set
Description: Clinical cure was defined as improvement in baseline signs and symptoms such that after study treatment, no further antimicrobial treatment for the index infection (i.e., cIAI or HAP/VAP) was required. Additionally, for cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. Clinical cure was determined by the Independent Clinical Adjudication Committee. Percentage of participants with clinical cure by pathogen resistance type (ATM non-susceptible and Meropenem non-susceptible based on European Committee on Antimicrobial Susceptibility Testing [EUCAST] criteria and Clinical and Laboratory Standards Institute [CLSI] criteria, Extended spectrum beta-lactamases [ESBL]-positive, Carbapenemase-positive, Serene Carbapenemase and Metallo-beta-lactamase-positive) is reported in this outcome measure.
Time Frame: At EOT visit (Within 24 hours after last infusion on Day 14)
Population: Micro-ITT analysis set was a subset of the ITT analysis set and included all participants who had at least one Gram-negative baseline pathogen from an adequate specimen obtained prior to the start of study treatment. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for specified rows.
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 177 | 94
Percentage of participants
  ATM non-susceptible, EUCAST: number analyzed (Participants) | 55 | 36
  ATM non-susceptible, EUCAST | 74.5 | 75.0
  ATM non-susceptible, CLSI: number analyzed (Participants) | 38 | 31
  ATM non-susceptible, CLSI | 68.4 | 74.2
  Meropenem non-susceptible, EUCAST: number analyzed (Participants) | 19 | 11
  Meropenem non-susceptible, EUCAST | 57.9 | 72.7
  Meropenem non-susceptible, CLSI: number analyzed (Participants) | 17 | 12
  Meropenem non-susceptible, CLSI | 58.8 | 75.0
  ESBL-positive: number analyzed (Participants) | 25 | 20
  ESBL-positive | 72.0 | 75.0
  Carbapenemase-positive: number analyzed (Participants) | 13 | 6
  Carbapenemase-positive | 61.5 | 50.0
  Serene Carbapenemase: number analyzed (Participants) | 7 | 3
  Serene Carbapenemase | 57.1 | 33.3
  Metallo-beta-lactamase-positive: number analyzed (Participants) | 7 | 3
  Metallo-beta-lactamase-positive | 57.1 | 66.7

40. Other Pre Specified Outcome: Percentage of Participants With Clinical Cure by Pathogen Resistance Type at TOC Visit: Micro-ITT Analysis Set
Description: Clinical cure was defined as improvement in baseline signs and symptoms such that after study treatment, no further antimicrobial treatment for the index infection (i.e., cIAI or HAP/VAP) was required. Additionally, for cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. Clinical cure was determined by the Independent Clinical Adjudication Committee. Percentage of participants with clinical cure by pathogen resistance type (ATM non-susceptible and Meropenem non-susceptible based on EUCAST criteria and CLSI criteria, ESBL-positive, Carbapenemase-positive, Serene Carbapenemase and Metallo-beta-lactamase-positive) is reported in this outcome measure.
Time Frame: At TOC (Day 28)
Population: as for outcome 39
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 177 | 94
Percentage of participants
  ATM non-susceptible, EUCAST: number analyzed (Participants) | 55 | 36
  ATM non-susceptible, EUCAST | 63.6 | 55.6
  ATM non-susceptible, CLSI: number analyzed (Participants) | 38 | 31
  ATM non-susceptible, CLSI | 60.5 | 61.3
  Meropenem non-susceptible,: number analyzed (Participants) | 19 | 11
  Meropenem non-susceptible, | 42.1 | 45.5
  Meropenem non-susceptible, CLSI: number analyzed (Participants) | 17 | 12
  Meropenem non-susceptible, CLSI | 41.2 | 50.0
  ESBL-positive: number analyzed (Participants) | 25 | 20
  ESBL-positive | 68.0 | 70.0
  Carbapenemase-positive: number analyzed (Participants) | 13 | 6
  Carbapenemase-positive | 30.8 | 33.3
  Serene Carbapenemase: number analyzed (Participants) | 7 | 3
  Serene Carbapenemase | 28.6 | 0
  Metallo-beta-lactamase-positive: number analyzed (Participants) | 7 | 3
  Metallo-beta-lactamase-positive | 28.6 | 66.7

41. Other Pre Specified Outcome: Percentage of Participants With Clinical Cure by Pathogen Resistance Type at EOT Visit: ME Analysis Set
Description: as for outcome 40
Time Frame: At EOT (Within 24 hours after last infusion on Day 14)
Population: The ME analysis set included all participants commonly included in both micro-ITT and CE analysis sets and included participants who had at least 1 etiologic pathogen from an adequate baseline culture regardless of susceptibility to study agents. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for specified rows.
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 149 | 79
Percentage of participants
  ATM non-susceptible, EUCAST: number analyzed (Participants) | 37 | 28
  ATM non-susceptible, EUCAST | 81.1 | 78.6
  ATM non-susceptible, CLSI: number analyzed (Participants) | 30 | 25
  ATM non-susceptible, CLSI | 76.7 | 76.0
  Meropenem non-susceptible, EUCAST: number analyzed (Participants) | 13 | 8
  Meropenem non-susceptible, EUCAST | 69.2 | 62.5
  Meropenem non-susceptible, CLSI: number analyzed (Participants) | 13 | 8
  Meropenem non-susceptible, CLSI | 69.2 | 62.5
  ESBL-positive: number analyzed (Participants) | 22 | 17
  ESBL-positive | 77.3 | 82.4
  Carbapenemase-positive: number analyzed (Participants) | 10 | 4
  Carbapenemase-positive | 80.0 | 25.0
  Serene Carbapenemase: number analyzed (Participants) | 6 | 3
  Serene Carbapenemase | 66.7 | 33.3
  Metallo-beta-lactamase-positive: number analyzed (Participants) | 4 | 1
  Metallo-beta-lactamase-positive | 100.0 | 0

42. Other Pre Specified Outcome: Percentage of Participants With Clinical Cure by Pathogen Resistance Type at TOC Visit: ME Analysis Set
Description: as for outcome 40
Time Frame: At TOC visit (Day 28)
Population: as for outcome 41
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 149 | 79
Percentage of participants
  ATM non-susceptible, EUCAST Criteria: number analyzed (Participants) | 37 | 28
  ATM non-susceptible, EUCAST Criteria | 70.3 | 60.7
  ATM non-susceptible, CLSI Criteria: number analyzed (Participants) | 30 | 25
  ATM non-susceptible, CLSI Criteria | 66.7 | 64.0
  Meropenem non-susceptible, EUCAST Criteria: number analyzed (Participants) | 13 | 8
  Meropenem non-susceptible, EUCAST Criteria | 46.2 | 37.5
  Meropenem non-susceptible, CLSI Criteria: number analyzed (Participants) | 13 | 8
  Meropenem non-susceptible, CLSI Criteria | 46.2 | 37.5
  ESBL-positive: number analyzed (Participants) | 22 | 17
  ESBL-positive | 72.7 | 76.5
  Carbapenemase-positive: number analyzed (Participants) | 10 | 4
  Carbapenemase-positive | 40.0 | 0
  Serene Carbapenemase: number analyzed (Participants) | 6 | 3
  Serene Carbapenemase | 33.3 | 0
  Metallo-beta-lactamase-positive: number analyzed (Participants) | 4 | 1
  Metallo-beta-lactamase-positive | 50.0 | 0

43. Other Pre Specified Outcome: Percentage of Participants With Favorable Per Participant Microbiological Response at EOT Visit: Micro-ITT Analysis Set
Description: as for outcome 9
Time Frame: At EOT visit (Within 24 hours after last infusion on Day 14)
Population: Micro-ITT analysis set is a subset of the ITT analysis set and included all participants who had at least one Gram-negative baseline pathogen from an adequate specimen obtained prior to the start of study treatment. Participants with a per participant response of indeterminate were excluded from this analysis. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 169 | 93
Percentage of participants | 84.6 | 83.9

44. Other Pre Specified Outcome: Percentage of Participants With Favorable Per Participant Microbiological Response at EOT Visit : ME Analysis Set
Description: as for outcome 9
Time Frame: At EOT visit (Within 24 hours after last infusion on Day 14)
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 149 | 79
Percentage of participants | 85.9 | 86.1

45. Other Pre Specified Outcome: Number of Participants With Favorable Microbiological Response Per-Pathogen at EOT Visit: Micro-ITT Analysis Set
Description: Participants were determined to have a favorable microbiological response if all baseline pathogens for that participant had a favorable outcome (eradicated or presumed eradicated). Eradication: Absence of causative pathogen from an appropriately obtained specimen at the site of infection. Presumed eradication: repeat culture of specimens were not performed/clinically indicated in a participant who had a clinical response of cure. Only those pathogens are reported which had more than or equal to 10 isolates for either treatment group.
Time Frame: At EOT (Within 24 hours after last infusion on Day 14)
Population: Micro-ITT analysis set is a subset of the ITT analysis set and included all participants who had at least one Gram-negative baseline pathogen from an adequate specimen obtained prior to the start of study treatment. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 177 | 94
Participants
  Escherichia coli: number analyzed (Participants) | 114 | 58
  Escherichia coli | 95 | 48
  Klebsiella pneumoniae: number analyzed (Participants) | 27 | 23
  Klebsiella pneumoniae | 19 | 18
  Pseudomonas aeruginosa: number analyzed (Participants) | 18 | 6
  Pseudomonas aeruginosa | 14 | 5
  Streptococcus anginosus group: number analyzed (Participants) | 17 | 6
  Streptococcus anginosus group | 13 | 4
  Bacteroides fragilis: number analyzed (Participants) | 16 | 9
  Bacteroides fragilis | 13 | 7
  Bacteroides thetaiotaomicron: number analyzed (Participants) | 11 | 1
  Bacteroides thetaiotaomicron | 8 | 1

46. Other Pre Specified Outcome: Number of Participants With Favorable Microbiological Response Per-Pathogen at at TOC Visit: Micro-ITT Analysis Set
Description: as for outcome 45
Time Frame: At TOC visit (Day 28)
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 177 | 94
Participants
  Escherichia coli: number analyzed (Participants) | 114 | 58
  Escherichia coli | 91 | 44
  Klebsiella pneumoniae: number analyzed (Participants) | 27 | 23
  Klebsiella pneumoniae | 14 | 15
  Pseudomonas aeruginosa: number analyzed (Participants) | 18 | 6
  Pseudomonas aeruginosa | 12 | 3
  Streptococcus anginosus group: number analyzed (Participants) | 17 | 6
  Streptococcus anginosus group | 12 | 4
  Bacteroides fragilis: number analyzed (Participants) | 16 | 9
  Bacteroides fragilis | 14 | 7
  Bacteroides thetaiotaomicron: number analyzed (Participants) | 11 | 1
  Bacteroides thetaiotaomicron | 8 | 1

47. Other Pre Specified Outcome: Number of Participants With Favorable Microbiological Response Per-Pathogen at EOT Visit: ME Analysis Set
Description: as for outcome 45
Time Frame: At EOT (Within 24 hours after last infusion on Day 14)
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 149 | 79
Participants
  Escherichia coli: number analyzed (Participants) | 101 | 53
  Escherichia coli | 90 | 44
  Klebsiella pneumoniae: number analyzed (Participants) | 23 | 20
  Klebsiella pneumoniae | 17 | 17
  Streptococcus anginosus group: number analyzed (Participants) | 14 | 5
  Streptococcus anginosus group | 13 | 3
  Bacteroides fragilis: number analyzed (Participants) | 15 | 8
  Bacteroides fragilis | 13 | 6
  Bacteroides thetaiotaomicron: number analyzed (Participants) | 11 | 1
  Bacteroides thetaiotaomicron | 8 | 1

48. Other Pre Specified Outcome: Number of Participants With Favorable Microbiological Response Per-Pathogen at TOC Visit: ME Analysis Set
Description: as for outcome 45
Time Frame: At TOC visit (Day 28)
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 149 | 79
Participants
  Escherichia coli: number analyzed (Participants) | 101 | 53
  Escherichia coli | 86 | 40
  Klebsiella pneumoniae: number analyzed (Participants) | 23 | 20
  Klebsiella pneumoniae | 13 | 14
  Streptococcus anginosus group: number analyzed (Participants) | 14 | 5
  Streptococcus anginosus group | 12 | 3
  Bacteroides fragilis: number analyzed (Participants) | 15 | 8
  Bacteroides fragilis | 14 | 6
  Bacteroides thetaiotaomicron: number analyzed (Participants) | 11 | 1
  Bacteroides thetaiotaomicron | 8 | 1

49. Other Pre Specified Outcome: Percentage of Participants With Favorable Per-Participant Microbiological Response by Pathogen Resistance Type at EOT Visit: Micro-ITT Analysis Set
Description: Participants were determined to have a favorable microbiological response if all baseline pathogens for that participant had a favorable outcome (eradicated or presumed eradicated). Eradication: Absence of causative pathogen from an appropriately obtained specimen at the site of infection. Presumed eradication: repeat culture of specimens were not performed/clinically indicated in a participant who had a clinical response of cure. Percentage of participants with favorable microbiological response by pathogen resistance type (ATM non-susceptible and Meropenem non-susceptible based on EUCAST criteria and CLSI criteria, ESBL-positive, Carbapenemase-positive, Serene Carbapenemase and Metallo-beta-lactamase-positive) is reported in this outcome measure.
Time Frame: At EOT (Within 24 hours after last infusion on Day 14)
Population: Micro-ITT analysis set=subset of ITT analysis set & included all participants who had at least 1 Gram-negative baseline pathogen from an adequate specimen obtained prior to start of study treatment.Here, 'Overall Number of Participants Analyzed' signifies participants included in micro-ITT analysis set and contributed data to table. Number Analyzed=number of participants evaluable for specified rows and participants with per participant response of indeterminate were excluded from analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 177 | 94
Percentage of participants
  ATM non-susceptible: CLSI: number analyzed (Participants) | 32 | 28
  ATM non-susceptible: CLSI | 68.8 | 78.6
  ATM non-susceptible : EUCAST: number analyzed (Participants) | 42 | 31
  ATM non-susceptible : EUCAST | 76.2 | 80.6
  Meropenem non-susceptible : CLSI: number analyzed (Participants) | 14 | 9
  Meropenem non-susceptible : CLSI | 57.1 | 66.7
  Meropenem non-susceptible : EUCAST: number analyzed (Participants) | 14 | 9
  Meropenem non-susceptible : EUCAST | 57.1 | 66.7
  ESBL-positive: number analyzed (Participants) | 23 | 19
  ESBL-positive | 78.3 | 84.2
  Carbapenamase-positive: number analyzed (Participants) | 10 | 4
  Carbapenamase-positive | 50.0 | 25.0
  Serene Carbapenamase-positive: number analyzed (Participants) | 6 | 3
  Serene Carbapenamase-positive | 33.3 | 33.3
  Metallo-beta-lactamase-positive: number analyzed (Participants) | 4 | 1
  Metallo-beta-lactamase-positive | 75.0 | 0.0

50. Other Pre Specified Outcome: Percentage of Participants With Favorable Per-Participant Microbiological Response by Pathogen Resistance Type at TOC Visit: Micro-ITT Analysis Set
Description: as for outcome 49
Time Frame: At TOC visit (Day 28)
Population: Micro-ITT analysis set=subset of ITT analysis set & included all participants who had at least 1 Gram-negative baseline pathogen from an adequate specimen obtained prior to start of study treatment. Here, 'Overall Number of Participants Analyzed' signifies participants included in micro-ITT analysis set and contributed data to table. Number Analyzed=number of participants evaluable for specified rows and participants with per participant response of indeterminate were excluded from analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 177 | 94
Percentage of participants
  ATM non-susceptible: CLSI: number analyzed (Participants) | 32 | 27
  ATM non-susceptible: CLSI | 59.4 | 59.3
  ATM non-susceptible: EUCAST: number analyzed (Participants) | 42 | 30
  ATM non-susceptible: EUCAST | 66.7 | 60.0
  Meropenem non-susceptible: CLSI: number analyzed (Participants) | 14 | 8
  Meropenem non-susceptible: CLSI | 28.6 | 25.0
  Meropenem non-susceptible : EUCAST: number analyzed (Participants) | 14 | 8
  Meropenem non-susceptible : EUCAST | 28.6 | 25.0
  ESBL-positive: number analyzed (Participants) | 23 | 19
  ESBL-positive | 73.9 | 73.7
  Carbapenamase-positive: number analyzed (Participants) | 10 | 4
  Carbapenamase-positive | 20.0 | 0.0
  Serene Carbapenamase-positive: number analyzed (Participants) | 6 | 3
  Serene Carbapenamase-positive | 16.7 | 0.0
  Metallo-beta-lactamase-positive: number analyzed (Participants) | 4 | 1
  Metallo-beta-lactamase-positive | 25.0 | 0.0

51. Other Pre Specified Outcome: Percentage of Participants With Favorable Per-Participant Microbiological Response by Pathogen Resistance Type at EOT Visit: ME Analysis Set
Description: Participants were determined to have a favorable microbiological response if all baseline pathogens for that participant had a favorable outcome (eradicated or presumed eradicated). Eradication: Absence of causative pathogen from an appropriately obtained specimen at the site of infection. Presumed eradication: repeat culture of specimens were not performed/clinically indicated in a participant who had a clinical response of cure. Percentage of participants with favorable microbiological response by pathogen resistance type (ATM non-susceptible, Meropenem non-susceptible based on EUCAST criteria and CLSI criteria, ESBL-positive, Carbapenemase-positive, Serene Carbapenemase and Metallo-beta-lactamase-positive) is reported in this outcome measure.
Time Frame: At EOT (Within 24 hours after last infusion on Day 14)
Population: ME analysis set =all participants commonly included in both micro-ITT and CE analysis sets and included participants who had at least 1 etiologic pathogen from an adequate baseline culture regardless of susceptibility to study agents. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for specified rows.
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 149 | 79
Percentage of participants
  ATM non-susceptible: CLSI: number analyzed (Participants) | 30 | 25
  ATM non-susceptible: CLSI | 70.0 | 80.0
  ATM non-susceptible: EUCAST: number analyzed (Participants) | 36 | 28
  ATM non-susceptible: EUCAST | 75.0 | 82.1
  Meropenem non-susceptible: CLSI: number analyzed (Participants) | 13 | 8
  Meropenem non-susceptible: CLSI | 53.8 | 62.5
  Meropenem non-susceptible: EUCAST: number analyzed (Participants) | 13 | 8
  Meropenem non-susceptible: EUCAST | 53.8 | 62.5
  ESBL-positive: number analyzed (Participants) | 22 | 17
  ESBL-positive | 77.3 | 88.2
  Carbapenamase-positive: number analyzed (Participants) | 9 | 4
  Carbapenamase-positive | 44.4 | 25.0
  Serene Carbapenamase-positive: number analyzed (Participants) | 6 | 3
  Serene Carbapenamase-positive | 33.3 | 33.3
  Metallo-beta-lactamase-positive: number analyzed (Participants) | 3 | 1
  Metallo-beta-lactamase-positive | 66.7 | 0.0

52. Other Pre Specified Outcome: Percentage of Participants With Favorable Per-Participant Microbiological Response by Pathogen Resistance Type at TOC Visit: ME Analysis Set
Description: as for outcome 51
Time Frame: At TOC visit (Day 28)
Population: as for outcome 51
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 149 | 79
Percentage of participants
  ATM non-susceptible: CLSI: number analyzed (Participants) | 30 | 25
  ATM non-susceptible: CLSI | 60.0 | 60.0
  ATM non-susceptible: EUCAST: number analyzed (Participants) | 36 | 28
  ATM non-susceptible: EUCAST | 66.7 | 60.7
  Meropenem non-susceptible: CLSI: number analyzed (Participants) | 13 | 8
  Meropenem non-susceptible: CLSI | 30.8 | 25.0
  Meropenem non-susceptible: EUCAST: number analyzed (Participants) | 13 | 8
  Meropenem non-susceptible: EUCAST | 30.8 | 25.0
  ESBL-positive: number analyzed (Participants) | 22 | 17
  ESBL-positive | 72.7 | 76.5
  Carbapenamase-positive: number analyzed (Participants) | 9 | 4
  Carbapenamase-positive | 22.2 | 0.0
  Serene Carbapenamase-positive: number analyzed (Participants) | 6 | 3
  Serene Carbapenamase-positive | 16.7 | 0.0
  Metallo-beta-lactamase-positive: number analyzed (Participants) | 3 | 1
  Metallo-beta-lactamase-positive | 33.3 | 0.0

53. Other Pre Specified Outcome: Percentage of Participants With Favorable Per-Pathogen Microbiological Response by Pathogen Resistance Type at EOT Visit: Micro-ITT Analysis Set
Description: Participants were determined to have a favorable microbiological response if all baseline pathogens for that participant had a favorable outcome (eradicated or presumed eradicated). Eradication: Absence of causative pathogen from an appropriately obtained specimen at the site of infection. Presumed eradication: repeat culture of specimens were not performed/clinically indicated in a participant who had a clinical response of cure. Percentage of participants with favorable per-pathogen microbiological response by pathogen resistance type (ATM non-susceptible, Meropenem non-susceptible based on EUCAST criteria and CLSI criteria, ESBL-positive, Carbapenemase-positive, Serene Carbapenemase and Metallo-beta-lactamase-positive) is reported in this outcome measure.
Time Frame: At EOT (Within 24 hours after last infusion on Day 14)
Population: as for outcome 45
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 177 | 94
Percentage of participants
  ATM non-susceptible: CLSI: number analyzed (Participants) | 41 | 31
  ATM non-susceptible: CLSI | 68.3 | 77.4
  ATM non-susceptible: EUCAST: number analyzed (Participants) | 60 | 37
  ATM non-susceptible: EUCAST | 73.3 | 78.4
  Meropenem non-susceptible: CLSI: number analyzed (Participants) | 20 | 12
  Meropenem non-susceptible: CLSI | 60.0 | 75.0
  Meropenem non-susceptible : EUCAST: number analyzed (Participants) | 22 | 11
  Meropenem non-susceptible : EUCAST | 59.1 | 72.7
  ESBL-positive: number analyzed (Participants) | 25 | 20
  ESBL-positive | 72.0 | 80.0
  Carbapenemase-positive: number analyzed (Participants) | 13 | 6
  Carbapenemase-positive | 61.5 | 50.0
  Serine-carbapenemase-positive: number analyzed (Participants) | 7 | 3
  Serine-carbapenemase-positive | 42.9 | 33.3
  Metallo-beta-lactamase-positive: number analyzed (Participants) | 7 | 3
  Metallo-beta-lactamase-positive | 71.4 | 66.7

54. Other Pre Specified Outcome: Percentage of Participants With Favorable Per-Pathogen Microbiological Response by Pathogen Resistance Type at TOC Visit: Micro-ITT Analysis Set
Description: as for outcome 53
Time Frame: At TOC visit (Day 28)
Population: as for outcome 45
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 177 | 94
Percentage of participants
  ATM non-susceptible: CLSI: number analyzed (Participants) | 41 | 31
  ATM non-susceptible: CLSI | 58.5 | 58.1
  ATM non-susceptible: EUCAST: number analyzed (Participants) | 60 | 37
  ATM non-susceptible: EUCAST | 63.3 | 56.8
  Meropenem non-susceptible: CLSI: number analyzed (Participants) | 20 | 12
  Meropenem non-susceptible: CLSI | 30.0 | 41.7
  Meropenem non-susceptible: EUCAST: number analyzed (Participants) | 22 | 11
  Meropenem non-susceptible: EUCAST | 31.8 | 36.4
  ESBL-positive: number analyzed (Participants) | 25 | 20
  ESBL-positive | 72.0 | 70.0
  Carbapenemase-positive: number analyzed (Participants) | 13 | 6
  Carbapenemase-positive | 23.1 | 33.3
  Serine-carbapenemase-positive: number analyzed (Participants) | 7 | 3
  Serine-carbapenemase-positive | 14.3 | 0.0
  Metallo-beta-lactamase-positive: number analyzed (Participants) | 7 | 3
  Metallo-beta-lactamase-positive | 28.6 | 66.7

55. Other Pre Specified Outcome: Percentage of Participants With Favorable Per-Pathogen Microbiological Response by Pathogen Resistance Type at EOT Visit: ME Analysis Set
Description: as for outcome 53
Time Frame: At EOT (Within 24 hours after last infusion on Day 14)
Population: as for outcome 41
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 149 | 79
Percentage of participants
  ATM non-susceptible: CLSI: number analyzed (Participants) | 33 | 25
  ATM non-susceptible: CLSI | 75.8 | 80.0
  ATM non-susceptible: EUCAST: number analyzed (Participants) | 42 | 29
  ATM non-susceptible: EUCAST | 78.6 | 82.8
  Meropenem non-susceptible: CLSI: number analyzed (Participants) | 16 | 8
  Meropenem non-susceptible: CLSI | 62.5 | 62.5
  Meropenem non-susceptible: EUCAST: number analyzed (Participants) | 16 | 8
  Meropenem non-susceptible: EUCAST | 62.5 | 62.5
  ESBL-positive: number analyzed (Participants) | 22 | 17
  ESBL-positive | 77.3 | 88.2
  Carbapenemase-positive: number analyzed (Participants) | 10 | 4
  Carbapenemase-positive | 70.0 | 25.0
  Serine-carbapenemase-positive: number analyzed (Participants) | 6 | 3
  Serine-carbapenemase-positive | 50. | 33.3
  Metallo-beta-lactamase-positive: number analyzed (Participants) | 4 | 1
  Metallo-beta-lactamase-positive | 100.0 | 0.0

56. Other Pre Specified Outcome: Percentage of Participants With Favorable Per-Pathogen Microbiological Response by Pathogen Resistance Type at TOC Visit: ME Analysis Set
Description: as for outcome 53
Time Frame: At TOC visit (Day 28)
Population: as for outcome 41
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 149 | 79
Percentage of participants
  ATM non-susceptible: CLSI: number analyzed (Participants) | 33 | 25
  ATM non-susceptible: CLSI | 63.6 | 60.0
  ATM non-susceptible: EUCAST: number analyzed (Participants) | 42 | 29
  ATM non-susceptible: EUCAST | 66.7 | 62.1
  Meropenem non-susceptible: CLSI: number analyzed (Participants) | 16 | 8
  Meropenem non-susceptible: CLSI | 31.3 | 25.0
  Meropenem non-susceptible : EUCAST: number analyzed (Participants) | 16 | 8
  Meropenem non-susceptible : EUCAST | 31.3 | 25.0
  ESBL-positive:: number analyzed (Participants) | 22 | 17
  ESBL-positive: | 77.3 | 76.5
  Carbapenemase-positive:: number analyzed (Participants) | 10 | 4
  Carbapenemase-positive: | 30.0 | 0.0
  Serine-carbapenemase-positive: number analyzed (Participants) | 6 | 3
  Serine-carbapenemase-positive | 16.7 | 0.0
  Metallo-beta-lactamase-positive:: number analyzed (Participants) | 4 | 1
  Metallo-beta-lactamase-positive: | 50.0 | 0.0

57. Other Pre Specified Outcome: Number of Participants According to Total Score for the Composite Endpoint of Symptom-Based Objective Clinical Measures: ITT Analysis Set
Time Frame: Up to Day 28
Population: The ITT analysis set included all randomized participants regardless of receipt of study drug. A composite scoring system was never developed and therefore there is no data to report for this outcome measure.
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 0 | 0

58. Other Pre Specified Outcome: Number of Participants According to Total Score for the Composite Endpoint of Symptom-Based Objective Clinical Measures: CE Analysis Set
Description: CE analysis set: all participants in ITT analysis set; met criteria for cIAI, or HAP/VAP; received at least 48 hours of study treatment or <48 hours of treatment before discontinuing study drug due to AE; no concomitant antibiotics for any baseline pathogens between first dose and TOC (except protocol-allowed antibiotics); no prior antibiotics other than allowed per protocol; no important protocol deviations; no clinical outcome of indeterminate at TOC; no monomicrobial infections due to non-eligible pathogens and did not have only Gram-positive pathogens.
Time Frame: Up to Day 28
Population: CE analysis set. A composite scoring system was never developed and therefore there is no data to report for this outcome measure.
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 0 | 0

59. Other Pre Specified Outcome: Percentage of Participants Who Died on or Before 14 Days From Randomization: ITT Analysis Set
Description: Percentage of participants who died on or before 14 days from randomization is reported in this outcome measure.
Time Frame: From randomization up to 14 days
Population: The ITT analysis set included all randomized participants regardless of receipt of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 282 | 140
Percentage of participants | 2.8 | 3.6

60. Other Pre Specified Outcome: Total Length of Hospital Stay up to TOC Visit: ITT Analysis Set
Description: The total length of hospital stay was defined as the total number of calendar days on which the participant was in the hospital from the date of randomization up to and including the specified time point of TOC.
Time Frame: From randomization up to Day 28
Population: The ITT analysis set included all randomized participants regardless of receipt of study drug. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 281 | 139
Days | 13.6 (9.42) | 12.9 (8.05)

61. Other Pre Specified Outcome: Total Length of Hospital Stay up to TOC Visit: CE Analysis Set
Description: The total length of hospital stay was defined as the total number of calendar days on which the participant was in the hospital from the date of randomization up to and including the specified time point of TOC. CE analysis set: all participants in ITT analysis set; met criteria for cIAI, or HAP/VAP; received at least 48 hours of study treatment or <48 hours of treatment before discontinuing study drug due to AE; no concomitant antibiotics for any baseline pathogens between first dose and TOC (except protocol-allowed antibiotics); no prior antibiotics other than allowed per protocol; no important protocol deviations; no clinical outcome of indeterminate at TOC; no monomicrobial infections due to non-eligible pathogens and did not have only Gram-positive pathogens.
Time Frame: From randomization up to Day 28
Population: CE analysis set.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 213 | 105
Days | 13.0 (8.55) | 12.3 (7.29)

62. Other Pre Specified Outcome: Duration of Study Treatment
Description: The duration of therapy in calendar days were calculated as follows: Date of last dose of study drug - date of first dose of study drug +1.
Time Frame: From first dose of study treatment until last dose of treatment (Up to 14 days)
Population: The safety analysis set included all participants who received any amount of study treatment.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 275 | 137
Days | 8.5 (3.52) | 8.9 (3.17)

63. Other Pre Specified Outcome: Length of Intensive Care Unit (ICU) Stay: ITT Analysis Set
Description: The total length of ICU stay was defined as the total number of calendar days on which the participant was in ICU for the period from date of randomization until the TOC visit.
Time Frame: From randomization until TOC visit (Up to Day 28)
Population: as for outcome 60
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 80 | 39
Days | 11.6 (9.10) | 12.5 (9.45)

64. Other Pre Specified Outcome: Length of Intensive Care Unit (ICU) Stay: CE Analysis Set
Description: The total length of ICU stay was defined as the total number of calendar days on which the participant was in ICU for the period from date of randomization until the TOC visit. CE analysis set: all participants in ITT analysis set; met criteria for cIAI, or HAP/VAP; received at least 48 hours of study treatment or <48 hours of treatment before discontinuing study drug due to AE; no concomitant antibiotics for any baseline pathogens between first dose and TOC (except protocol-allowed antibiotics); no prior antibiotics other than allowed per protocol; no important protocol deviations; no clinical outcome of indeterminate at TOC; no monomicrobial infections due to non-eligible pathogens and did not have only Gram-positive pathogens.
Time Frame: From randomization until TOC visit (Up to Day 28)
Population: CE analysis set. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 54 | 24
Days | 12.1 (9.23) | 12.4 (9.38)

65. Other Pre Specified Outcome: Number of Participants Admitted to the ICU: ITT Analysis Set
Description: Number of participants admitted to the ICU up to TOC were reported in this outcome measure.
Time Frame: From randomization until TOC visit (Up to Day 28)
Population: The ITT analysis set included all randomized participants regardless of receipt of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 282 | 140
Participants | 80 | 39

66. Other Pre Specified Outcome: Number of Participants Admitted to the ICU: CE Analysis Set
Description: The number of participants admitted to the ICU were reported in this outcome measure. CE analysis set: all participants in ITT analysis set; met criteria for cIAI, or HAP/VAP; received at least 48 hours of study treatment or <48 hours of treatment before discontinuing study drug due to AE; no concomitant antibiotics for any baseline pathogens between first dose and TOC (except protocol-allowed antibiotics); no prior antibiotics other than allowed per protocol; no important protocol deviations; no clinical outcome of indeterminate at TOC; no monomicrobial infections due to non-eligible pathogens and did not have only Gram-positive pathogens.
Time Frame: From randomization until TOC visit (Up to Day 28)
Population: CE analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 213 | 105
Participants | 54 | 24

67. Other Pre Specified Outcome: Number of Participants With Mechanical Ventilation: ITT Analysis Set
Description: Number of participants with mechanical ventilation were reported in this outcome measure.
Time Frame: From randomization until TOC visit (Up to Day 28)
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 74 | 36
Participants | 43 | 21

68. Other Pre Specified Outcome: Number of Participants With Mechanical Ventilation: CE Analysis Set
Description: Number of participants with mechanical ventilation were reported in this outcome measure. CE analysis set: all participants in ITT analysis set; met criteria for cIAI, or HAP/VAP; received at least 48 hours of study treatment or <48 hours of treatment before discontinuing study drug due to AE; no concomitant antibiotics for any baseline pathogens between first dose and TOC (except protocol-allowed antibiotics); no prior antibiotics other than allowed per protocol; no important protocol deviations; no clinical outcome of indeterminate at TOC; no monomicrobial infections due to non-eligible pathogens and did not have only Gram-positive pathogens.
Time Frame: From randomization until TOC visit (Up to Day 28)
Population: as for outcome 64
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 45 | 22
Participants | 24 | 13

69. Other Pre Specified Outcome: Duration of Mechanical Ventilation in HAP/VAP Participants: ITT Analysis Set
Description: Duration of mechanical ventilation was defined as the total number of calendar days on which the participant required mechanical ventilation from the date of randomization up to TOC.
Time Frame: From randomization until TOC visit (Up to Day 28)
Population: as for outcome 60
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 43 | 21
Days | 14.2 (9.94) | 16.7 (11.16)

70. Other Pre Specified Outcome: Duration of Mechanical Ventilation in HAP/VAP Participants: CE Analysis Set
Description: Duration of mechanical ventilation was defined as the total number of calendar days on which the participant required mechanical ventilation from the date of randomization up to TOC. CE analysis set: all participants in ITT analysis set; met criteria for cIAI, or HAP/VAP; received at least 48 hours of study treatment or <48 hours of treatment before discontinuing study drug due to AE; no concomitant antibiotics for any baseline pathogens between first dose and TOC (except protocol-allowed antibiotics); no prior antibiotics other than allowed per protocol; no important protocol deviations; no clinical outcome of indeterminate at TOC; no monomicrobial infections due to non-eligible pathogens and did not have only Gram-positive pathogens.
Time Frame: From randomization until TOC visit (Up to Day 28)
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 24 | 13
Days | 17.4 (8.99) | 19.5 (11.16)

71. Other Pre Specified Outcome: Number of Participants With Unplanned Surgical Interventions in Complicated Intra-abdominal Infections (cIAI) Participants: ITT Analysis Set
Description: Unplanned surgical interventions was defined as those occurring after the initial qualifying surgical intervention and prior to the TOC visit. Number of cIAI participants with unplanned surgical intervention according to clinical response categories of cure and failure is reported in this outcome measure.
Time Frame: From randomization until TOC visit (Up to Day 28)
Population: The ITT analysis set included all randomized participants regardless of receipt of study drug. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 193 | 100
Participants
  Cure: number analyzed (Participants) | 159 | 77
  Cure | 1 | 1
  Failure: number analyzed (Participants) | 34 | 23
  Failure | 5 | 10

72. Other Pre Specified Outcome: Number of Participants With Unplanned Surgical Interventions in cIAI Participants: CE Analysis Set
Description: as for outcome 71
Time Frame: From randomization until TOC visit (Up to Day 28)
Population: CE analysis set. All participants reported under 'Overall Number of Participants Analyzed' include participants evaluable for this outcome measure and contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
Number analyzed (Participants) | 168 | 83
Participants
  Cure: number analyzed (Participants) | 143 | 66
  Cure | 1 | 1
  Failure: number analyzed (Participants) | 25 | 17
  Failure | 5 | 9

ADVERSE EVENTS:
Time Frame: All-cause mortality: From signing of informed consent until end of late follow up visit (Day 45); non-SAEs and SAEs: From start of study treatment until end of late follow-up visit (Up to Day 45).
Description: All-cause mortality is presented for ITT analysis set and non-SAEs and SAEs are presented for Safety analysis set.
Arm/Group | Aztreonam-avibactam ± Metronidazole | Meropenem± Colistimethate
All-Cause Mortality (participants affected / at risk) | 20/282 | 11/140
Serious Adverse Events (participants affected / at risk) | 53/275 | 25/137
Other Adverse Events (participants affected / at risk) | 113/275 | 45/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aztreonam-avibactam ± Metronidazole (N=275) | Meropenem± Colistimethate (N=137)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Myxomatous mitral valve degeneration (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 | 2
Melaena (Gastrointestinal disorders) | 0 | 1
Localised oedema (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 4 | 2
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abdominal wall infection (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 3 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 0
Central nervous system infection (Infections and infestations) | 0 | 1
Chronic hepatitis B (Infections and infestations) | 0 | 1
Device related bacteraemia (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 1
Pneumonia aspiration (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 2
Septic shock (Infections and infestations) | 2 | 3
Tracheobronchitis (Infections and infestations) | 1 | 0
Fat embolism (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain dislocation syndrome (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Device dislocation (Product Issues) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Convalescent (Social circumstances) | 0 | 1
Circulatory collapse (Vascular disorders) | 2 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aztreonam-avibactam ± Metronidazole (N=275) | Meropenem± Colistimethate (N=137)
Anaemia (Blood and lymphatic system disorders) | 20 | 7
Atrial fibrillation (Cardiac disorders) | 6 | 1
Abdominal distension (Gastrointestinal disorders) | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 6 | 4
Constipation (Gastrointestinal disorders) | 8 | 2
Diarrhoea (Gastrointestinal disorders) | 16 | 5
Nausea (Gastrointestinal disorders) | 10 | 3
Vomiting (Gastrointestinal disorders) | 10 | 2
Injection site reaction (General disorders) | 1 | 4
Pyrexia (General disorders) | 14 | 5
Hepatic function abnormal (Hepatobiliary disorders) | 11 | 3
Hypertransaminasaemia (Hepatobiliary disorders) | 6 | 1
Alanine aminotransferase increased (Investigations) | 18 | 7
Aspartate aminotransferase increased (Investigations) | 15 | 5
Blood alkaline phosphatase increased (Investigations) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 16 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 0
Hypertension (Vascular disorders) | 5 | 3
Phlebitis (Vascular disorders) | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT03329092/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT03329092/SAP_001.pdf